CLINICAL TRIAL: NCT03284710
Title: A Phase 1/2a Partially Double-blinded, Randomized Clinical Trial to Characterize the Safety and Immunogenicity of Clade C ALVAC-HIV (vCP2438) and Bivalent Subtype C gp120 Alone, With MF59 Adjuvant, and With Alum Adjuvant in Healthy, HIV-uninfected Adult Participants
Brief Title: Safety and Immunogenicity of Clade C ALVAC and gp120 HIV Vaccine
Acronym: HVTN107
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); Sanofi Pasteur, a Sanofi Company (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 107
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: ALVAC-HIV + gp120/MF59 (Active Comparator): Participants will receive the ALVAC-HIV (vCP2438) vaccine in the left deltoid at months 0, 1, 3, 6, and 12, and Bivalent Subtype C gp120/MF59 in the right deltoid at months 3, 6, and 12. All injections are via needle and syringe.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent Subtype C gp120/MF59
- Group 2: ALVAC-HIV + gp120/Al(OH)3 (Active Comparator): Participants will receive the ALVAC-HIV (vCP2438) vaccine in the left deltoid at months 0, 1, 3, 6, and 12, and Bivalent Subtype C gp120 admixed with Al(OH)3 Suspension in the right deltoid at months 3, 6, and 12. All injections are via needle and syringe.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent Subtype C gp120 admixed with Al(OH)3 Suspension
- Group 3: ALVAC-HIV + gp120/MF59 (Active Comparator): Participants will receive the ALVAC-HIV (vCP2438) vaccine in the left deltoid and Bivalent Subtype C gp120/MF59 in the right deltoid at months 0, 1, 6, and 12. All injections are via needle and syringe.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent Subtype C gp120/MF59
- Group 4: ALVAC-HIV + gp120 (Active Comparator): Participants will receive the ALVAC-HIV (vCP2438) vaccine in the left deltoid at months 0, 1, 3, 6, and 12, and Bivalent Subtype C gp120 in the right deltoid at months 3, 6, and 12. All injections are via needle and syringe.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent Subtype C gp120

INTERVENTIONS:
Biological: ALVAC-HIV (vCP2438) — Expresses the gene products ZM96 gp120 (clade C strain) linked to the sequences encoding the HIV-1 transmembrane (TM) anchor sequence of gp41 (28 amino acids clade B LAI strain) and gag and pro (clade B LAI strain); formulated as a lyophilized vaccine for injection at a viral titer ≥ 1 × 10^6 cell culture infectious dose (CCID)50 and < 1 × 10^8 CCID50 (nominal dose of 10^7 CCID50) and reconstituted with 1mL of sterile sodium chloride solution (NaCl 0.4%) for intramuscular (IM) injection as a single dose
Biological: Bivalent Subtype C gp120/MF59 — Consists of 2 subtype C recombinant monomeric proteins, TV1.C gp120 Env and 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant (an oil-in-water emulsion); delivered as a 0.5 mL IM injection
  Arms: Group 1: ALVAC-HIV + gp120/MF59; Group 3: ALVAC-HIV + gp120/MF59
Biological: Bivalent Subtype C gp120 admixed with Al(OH)3 Suspension — Consists of 2 subtype C recombinant monomeric proteins, TV1.C gp120 Env and 1086.C gp120 Env, each at a dose of 100 mcg, admixed with Aluminum Hydroxide Suspension (~625 mcg aluminum content); delivered as a 0.5 mL IM injection
  Arms: Group 2: ALVAC-HIV + gp120/Al(OH)3
Biological: Bivalent Subtype C gp120 — Consists of 2 subtype C recombinant monomeric proteins, TV1.C gp120 Env and 1086.C gp120 Env, each at a dose of 100 mcg, mixed with sodium chloride for injection, 0.9%; delivered as a 0.5 mL IM injection
  Arms: Group 4: ALVAC-HIV + gp120

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to an HIV clade C vaccine and to an MF59- or alum-adjuvanted clade C Env protein in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity to vCP2438 (an HIV clade C vaccine) and to an unadjuvanted or MF59- or alum-adjuvanted bivalent clade C gp120 in healthy, HIV-uninfected adults.

The study will enroll healthy, HIV-uninfected participants aged 18 to 40 years. Participants will be randomly assigned to one of 4 groups. [describe further]

Study visits will include a physical examination, an interview and/or questionnaire, HIV testing and HIV risk-reduction counseling, and urine and blood collection. A subset of participants will provide rectal fluid, cervical fluid, semen, or stool samples.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

1. Age of 18 to 40 years
2. Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Agrees not to enroll in another study of an investigational research agent
6. Good general health as shown by medical history, physical exam, and screening laboratory tests

   HIV-Related Criteria:
7. Willingness to receive HIV test results
8. Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
9. Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

   Laboratory Inclusion Values

   Hemogram/Complete blood count (CBC)
10. Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
11. White blood cell count = 3,300 to 12,000 cells/mm^3
12. Total lymphocyte count ≥ 800 cells/mm^3
13. Remaining differential either within institutional normal range or with site physician approval
14. Platelets = 125,000 to 550,000/mm^3

    Chemistry
15. Chemistry panel: ALT, AST, and ALP < 1.25 times the institutional upper limit of normal; creatinine ≤ institutional upper limit of normal.

    Virology
16. Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
17. Negative Hepatitis B surface antigen (HBsAg)
18. Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive Urine
19. Normal urine:

    * Negative urine glucose, and
    * Negative or trace urine protein, and
    * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

    Reproductive Status
20. Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
21. Reproductive status: A volunteer who was born female must:

    * Agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using condoms (male or female), or diaphragm or cervical cap, PLUS 1 of the following methods: Intrauterine device (IUD), Hormonal contraception (in accordance with Republic of South Africa: National Contraception Clinical Guidelines), successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or any other contraceptive method approved by the HVTN 107 Protocol Safety Review Team
    * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
    * Or be sexually abstinent.
22. Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

    Other
23. Volunteers who were born female consenting to provide cervical samples: pap smear within the 3 years prior to enrollment, with the latest result reported as normal or ASCUS (atypical squamous cells of undetermined significance); for those 21 years and older that have not had a pap smear within the last 3 years prior to enrollment, must be willing to undergo a pap smear with the result reported as normal or ASCUS prior to sample collection.

Exclusion Criteria:

General

1. Blood products received within 120 days before first vaccination
2. Investigational research agents received within 30 days before first vaccination
3. Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
4. Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 107 study
5. Pregnant or breastfeeding

   Vaccines and other Injections
6. HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 107 PSRT will determine eligibility on a case-by-case basis.
7. Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure in a volunteer's country of residence. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 107 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 107 PSRT on a case-by-case basis.
8. Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
9. Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
10. Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

    Immune System
11. Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.)
12. Serious adverse reactions to vaccines or to vaccine components such as eggs, egg products, or neomycin, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
13. Immunoglobulin received within 60 days before first vaccination
14. Autoimmune disease
15. Immunodeficiency

    Clinically significant medical conditions
16. Untreated or incompletely treated syphilis infection
17. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated injections or blood draws,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
    * Any condition specifically listed among the exclusion criteria below.
18. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
19. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
20. Current anti-tuberculosis (TB) prophylaxis or therapy
21. Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

    Exclude a volunteer who:
    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
    * Uses moderate/high dose inhaled corticosteroids, or
    * In the past year has either of the following:

      * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
      * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
22. Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
23. Thyroidectomy, or thyroid disease requiring medication during the last 12 months
24. Hypertension:

    * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
    * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
25. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
26. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
27. Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
28. Asplenia: any condition resulting in the absence of a functional spleen
29. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goepfert, Study Chair — University of Alabama at Birmingham; Kathy Mngadi, Study Chair — Centre for the AIDS Programme of Research in South Africa
Locations (6):
- Polana Canico Health Research and Training Center (CISPOC), National Institute of Health (INS) CRS, Maputo, Mozambique
- South Africa (4):
  - Aurum Tembisa CRS, Johannesburg, Gauteng
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - eThekwini CRS, Durban, KwaZulu-Natal
  - Emavundleni CRS, Cape Town, Western Cape
- Seke South CRS, Chitungwiza, Mashonaland East Province, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Moodie Z, Andersen-Nissen E, Grunenberg N, Dintwe OB, Omar FL, Kee JJ, Bekker LG, Laher F, Naicker N, Jani I, Mgodi NM, Hunidzarira P, Sebe M, Miner MD, Polakowski L, Ramirez S, Nebergall M, Takuva S, Sikhosana L, Heptinstall J, Seaton KE, De Rosa S, Diazgranados CA, Koutsoukos M, Van Der Meeren O, Barnett SW, Kanesa-Thasan N, Kublin JG, Tomaras GD, McElrath MJ, Corey L, Mngadi K, Goepfert P; HVTN 107 Protocol Team. Safety and immunogenicity of a subtype C ALVAC-HIV (vCP2438) vaccine prime plus bivalent subtype C gp120 vaccine boost adjuvanted with MF59 or alum in healthy adults without HIV (HVTN 107): A phase 1/2a randomized trial. PLoS Med. 2024 Mar 19;21(3):e1004360. doi: 10.1371/journal.pmed.1004360. eCollection 2024 Mar. PMID 38502656

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120/MF59 (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
- Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120 (an admixture of 100 mcg of TV1.C gp120 and 100 mcg of 1806.C gp120) admixed with Aluminum Hydroxide Suspension to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
- Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 6, and 12 AND Bivalent Subtype C gp120/MF59 (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 0, 1, 6, and 12
- Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120 (an admixture of 100 mcg of TV1.C gp120 and 100 mcg of 1806.C gp120) admixed with Sodium Chloride for Injection, 0.9% to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
Period: Overall Study
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Started | 36 | 36 | 36 | 24
Month 6.5 Immunogenicity Timepoint | 31 | 31 | 31 | 18
Month 12 Immunogenicity Timepoint | 30 | 31 | 31 | 17
Month 12.5 Immunogenicity Timepoint | 0 | 0 | 0 | 0
Month 18 Immunogenicity Timepoint | 0 | 0 | 0 | 0
Completed | 30 | 31 | 32 | 16
Not Completed | 6 | 5 | 4 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 6
Not completed — Lost to Follow-up | 3 | 3 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Participant Unable to Adhere to Visit Schedule | 1 | 0 | 0 | 1
Not completed — HIV Infection | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12) | Total
Number analyzed (Participants) | 36 | 36 | 36 | 24 | 132
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 39] | 25 [18 to 37] | 25 [19 to 39] | 25 [18 to 33] | 25 [18 to 39]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 7 | 4 | 4 | 6 | 21
  21 - 30 years | 24 | 28 | 29 | 16 | 97
  31 - 40 years | 5 | 4 | 3 | 2 | 14
  41 - 50 years | 0 | 0 | 0 | 0 | 0
  Above 50 years | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 20 | 15 | 79
  Male | 13 | 15 | 16 | 9 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 36 | 36 | 24 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 36 | 36 | 36 | 24 | 132
Region of Enrollment [Count of Participants; unit: Participants]
  Mozambique | 7 | 7 | 7 | 3 | 24
  South Africa | 21 | 21 | 21 | 17 | 80
  Zimbabwe | 8 | 8 | 8 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Vaccine-induced Systemic IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C) in Group 1 and Group 2
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if they meet three criteria: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI.
Time Frame: Measured at Month 6.5
Population: Overall Number of Participants Analyzed represents the HIV uninfected participants with specimens at Month 6.5. "Number Analyzed" shows the number of participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12)
Number analyzed (Participants) | 29 | 28
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 29 | 27
  1086C_D7gp120.avi/293F | 29 | 26
  96ZM651.D11gp120.avi: number analyzed (Participants) | 28 | 28
  96ZM651.D11gp120.avi | 27 | 27
  TV1c8_D11gp120.avi/293F | 29 | 27
Statistical Analysis 1: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to 1086C_D7gp120.avi/293F in Group 1 versus Group 2; Test type: Other; p = 0.358, Barnard's test — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to 96ZM651.D11gp120.avi in Group 1 versus Group 2; Test type: Other; p = 1.000, Barnard's test — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to TV1c8_D11gp120.avi/293F in Group 1 versus Group 2; Test type: Other; p = 0.361, Barnard's test — The threshold for statistical significance was p = 0.05

2. Primary Outcome: Level of Vaccine-induced Systemic IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C) in Group 1 and Group 2
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Comparisons were performed among positive responders only (positivity criteria are described in Outcome 1).
Time Frame: Measured at Month 6.5
Population: "Overall Number of Participants Analyzed" represents the HIV uninfected participants with specimens at Month 6.5. "Number Analyzed" shows the number of participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12)
Number analyzed (Participants) | 29 | 27
relative fluorescence units
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 29 | 26
  1086C_D7gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  96ZM651.D11gp120.avi: number analyzed (Participants) | 27 | 27
  96ZM651.D11gp120.avi | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  TV1c8_D11gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000]
Statistical Analysis 1: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to 1086C_D7gp120.avi/293F in Group 1 versus Group 2; Test type: Other; p = 0.238, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to 96ZM651.D11gp120.avi in Group 1 versus Group 2; Test type: Other; p = 0.893, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12); IgGAb binding to TV1c8_D11gp120.avi/293F in Group 1 versus Group 2; Test type: Other; p = 0.411, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05

3. Primary Outcome: Occurrence of Vaccine-induced Serum IgA Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C) in Group 1 and Group 3
Description: Serum IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:10 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if they meet three criteria: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI.
Time Frame: Measured at Month 6.5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12)
Number analyzed (Participants) | 26 | 30
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 24 | 29
  1086C_D7gp120.avi/293F | 22 | 27
  96ZM651.D11gp120.avi | 12 | 22
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 25 | 29
  TV1c8_D11gp120.avi/293F | 18 | 27
Statistical Analysis 1: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to 1086C_D7gp120.avi/293F in Group 1 versus Group 3; Test type: Other; p = 1.000, Barnard's test — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to 96ZM651.D11gp120.avi in Group 1 versus Group 3; Test type: Other; p = 0.044, Barnard's test — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to TV1c8_D11gp120.avi/293F in Group 1 versus Group 3; Test type: Other; p = 0.045, Barnard's test — The threshold for statistical significance was p = 0.05

4. Primary Outcome: Level of Vaccine-induced Serum IgA Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C) in Group 1 and Group 3
Description: Serum IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:10 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Comparisons were performed among positive responders only (positivity criteria are described in Outcome 1).
Time Frame: Measured at Month 6.5
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12)
Number analyzed (Participants) | 22 | 27
relative fluorescence units
  1086C_D7gp120.avi/293F | 22000 [17472 to 22000] | 22000 [22000 to 22000]
  96ZM651.D11gp120.avi: number analyzed (Participants) | 12 | 22
  96ZM651.D11gp120.avi | 8047.1 [6816.6 to 13252.6] | 7595.5 [5318.3 to 13822.1]
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 18 | 27
  TV1c8_D11gp120.avi/293F | 8312.8 [3759.4 to 19844.6] | 12210.8 [6345.9 to 22000]
Statistical Analysis 1: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to 1086C_D7gp120.avi/293F in Group 1 versus Group 3; Test type: Other; p = 0.215, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to 96ZM651.D11gp120.avi in Group 1 versus Group 3; Test type: Other; p = 0.683, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) vs Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12); IgAAb binding to TV1c8_D11gp120.avi/293F in Group 1 versus Group 3; Test type: Other; p = 0.322, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05

5. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at Months 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Pain: None | 21 | 20 | 22 | 17
  Pain: Mild | 14 | 13 | 13 | 7
  Pain: Moderate | 1 | 3 | 1 | 0
  Pain: Severe | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 20 | 20 | 25 | 16
  Tenderness: Mild | 16 | 15 | 11 | 8
  Tenderness: Moderate | 0 | 1 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 18 | 15 | 21 | 14
  Pain and/or Tenderness: Mild | 17 | 18 | 14 | 10
  Pain and/or Tenderness: Moderate | 1 | 3 | 1 | 0
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 5
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at Months 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Erythema: None | 30 | 31 | 33 | 22
  Erythema: Not gradable | 4 | 5 | 2 | 1
  Erythema: Mild | 1 | 0 | 1 | 1
  Erythema: Moderate | 1 | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0 | 0
  Erythema: Potentially Life-threatening | 0 | 0 | 0 | 0
  Induration: None | 29 | 28 | 34 | 19
  Induration: Not gradable | 2 | 7 | 2 | 2
  Induration: Mild | 1 | 0 | 0 | 2
  Induration: Moderate | 4 | 1 | 0 | 1
  Induration: Severe | 0 | 0 | 0 | 0
  Induration: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 28 | 27 | 32 | 18
  Erythema and/or Induration: Not gradable | 3 | 8 | 3 | 2
  Erythema and/or Induration: Mild | 1 | 0 | 1 | 3
  Erythema and/or Induration: Moderate | 4 | 1 | 0 | 1
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at Months 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Malaise and/or fatigue: None | 32 | 28 | 30 | 21
  Malaise and/or fatigue: Mild | 4 | 7 | 6 | 3
  Malaise and/or fatigue: Moderate | 0 | 1 | 0 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 36 | 35 | 35 | 22
  Myalgia: Mild | 0 | 1 | 1 | 2
  Myalgia: Moderate | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 28 | 28 | 29 | 19
  Headache: Mild | 8 | 6 | 7 | 5
  Headache: Moderate | 0 | 2 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 30 | 34 | 32 | 23
  Nausea: Mild | 6 | 2 | 4 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 36 | 35 | 36 | 24
  Vomiting: Mild | 0 | 1 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 36 | 34 | 33 | 23
  Chills: Mild | 0 | 2 | 3 | 1
  Chills: Moderate | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 34 | 34 | 34 | 24
  Arthralgia: Mild | 2 | 2 | 2 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 23 | 23 | 25 | 17
  Max. Systemic Symptoms: Mild | 13 | 11 | 11 | 7
  Max. Systemic Symptoms: Moderate | 0 | 2 | 0 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Temperature: None | 36 | 31 | 35 | 24
  Temperature: Mild | 0 | 3 | 1 | 0
  Temperature: Moderate | 0 | 1 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 1 | 0 | 0

8. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through 30 days after each vaccine dose at Months 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Related | 1 | 2 | 0 | 0
  Not Related | 27 | 26 | 26 | 15
  No AE Reported | 8 | 8 | 10 | 9

9. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: For participants reporting multiple AEs over the time frame, the maximum severity grade is counted.
Time Frame: Measured through 30 days after each vaccine dose at Months 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Mild | 5 | 7 | 12 | 2
  Moderate | 18 | 16 | 12 | 12
  Severe | 3 | 4 | 1 | 1
  Potentially Life-Threatening | 2 | 1 | 1 | 0
  Death | 0 | 0 | 0 | 0
  No AE Reported | 8 | 8 | 10 | 9

10. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Measured as outlined in Version 2.0 (January 2010) of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual).
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Yes | 1 | 0 | 0 | 1
  No | 27 | 28 | 26 | 14
  No AE Reported | 8 | 8 | 10 | 9

11. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: There were no adverse events of special interest reported by any participant.
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120/MF59® (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
- Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 6, and 12 AND Bivalent Subtype C gp120/MF59® (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 0, 1, 6, and 12
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants Reporting New Chronic Conditions (Requiring Medical Intervention for >= 30 Days)
Description: New chronic conditions are adverse events that require medical intervention for >= 30 days.
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Yes | 0 | 1 | 0 | 2
  No | 28 | 27 | 26 | 13
  No AE Reported | 8 | 8 | 10 | 9

13. Primary Outcome: Chemistry and Hematology Laboratory Measures - ALT (SGPT), AST, Alkaline Phosphatase
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, Days 7, 42, 98, 182, 378, and 455
Population: "Overall Number of Participants Analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
U/L
  Alkaline Phosphatase (U/L)- Screening | 72 [59 to 87] | 70 [62 to 89] | 76 [63.5 to 90.5] | 79.5 [65.5 to 94]
  Alkaline Phosphatase (U/L)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  Alkaline Phosphatase (U/L)- Day7 | 66.5 [58 to 83] | 68 [57 to 85] | 70 [62 to 82] | 75.5 [58 to 84]
  Alkaline Phosphatase (U/L)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Alkaline Phosphatase (U/L)- Day42 | 70 [57 to 84] | 71.5 [60 to 83] | 70.5 [62 to 90] | 78 [64 to 89]
  Alkaline Phosphatase (U/L)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Alkaline Phosphatase (U/L)- Day98 | 67.5 [60 to 79] | 64 [54 to 84] |  | 77 [62 to 87]
  Alkaline Phosphatase (U/L)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Alkaline Phosphatase (U/L)- Day182 | 70 [58 to 85] | 64 [56 to 78] | 70 [58 to 88] | 77.5 [61 to 84]
  Alkaline Phosphatase (U/L)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Alkaline Phosphatase (U/L)- Day378 | 70 [58.5 to 82.5] | 65 [54 to 83] | 73 [68 to 89] | 77.5 [55 to 95]
  Alkaline Phosphatase (U/L)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Alkaline Phosphatase (U/L)- Day455 | 71.5 [59 to 82] | 65 [54 to 81] | 71.5 [64 to 89.5] | 76.5 [66 to 89]
  AST (U/L)- Screening | 19 [16.5 to 22] | 20 [17.5 to 24] | 21.5 [19 to 24.5] | 17 [16.5 to 23]
  AST (U/L)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  AST (U/L)- Day7 | 18 [16.5 to 23] | 20 [17 to 22] | 21 [18 to 23] | 19 [16 to 20]
  AST (U/L)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  AST (U/L)- Day42 | 19 [15 to 25] | 21 [17 to 26] | 21 [18 to 24] | 21 [17 to 25]
  AST (U/L)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  AST (U/L)- Day98 | 21 [16 to 23.5] | 20 [17 to 27] |  | 20 [18 to 27]
  AST (U/L)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  AST (U/L)- Day182 | 20 [18 to 24] | 21 [18 to 25] | 21 [19 to 26] | 18.5 [16 to 26]
  AST (U/L)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  AST (U/L)- Day378 | 20 [16.5 to 27] | 19 [18 to 23] | 22 [19 to 29] | 21.5 [18 to 25]
  AST (U/L)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  AST (U/L)- Day455 | 22.5 [17 to 26] | 20 [17 to 24] | 21 [18.5 to 26] | 19 [16 to 27]
  ALT (SGPT) (U/L)- Screening | 15 [13 to 19] | 15 [11 to 20.5] | 16.5 [13.5 to 21.5] | 14.5 [12 to 20]
  ALT (SGPT) (U/L)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  ALT (SGPT) (U/L)- Day7 | 15.5 [12 to 19.5] | 16 [12 to 19] | 15 [11 to 19] | 15.5 [11 to 20]
  ALT (SGPT) (U/L)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  ALT (SGPT) (U/L)- Day42 | 16 [12 to 19] | 18.5 [11 to 25] | 15 [12 to 18] | 17.5 [12 to 22]
  ALT (SGPT) (U/L)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  ALT (SGPT) (U/L)- Day98 | 16 [13 to 20] | 15 [11 to 23] |  | 17 [12 to 19]
  ALT (SGPT) (U/L)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  ALT (SGPT) (U/L)- Day182 | 18 [13 to 20] | 16.5 [13 to 23] | 15 [12 to 23] | 15 [11 to 22]
  ALT (SGPT) (U/L)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  ALT (SGPT) (U/L)- Day378 | 16 [13 to 19.5] | 16 [11 to 24] | 15 [12 to 24] | 19 [12 to 24]
  ALT (SGPT) (U/L)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  ALT (SGPT) (U/L)- Day455 | 16 [14 to 20] | 16 [13 to 22] | 16 [11 to 21] | 15 [12 to 22]

14. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine
Description: as for outcome 13
Time Frame: Measured during screening, Days 7, 42, 98, 182, 378, and 455
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
g/dL
  Creatinine (g/dL)- Screening | 0.00071 [0.0006 to 0.00082] | 0.0007 [0.000605 to 0.000805] | 0.000705 [0.00061 to 0.00084] | 0.0007 [0.0006 to 0.0008]
  Creatinine (g/dL)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  Creatinine (g/dL)- Day7 | 0.00071 [0.000675 to 0.000845] | 0.0007 [0.0006 to 0.0008] | 0.0007 [0.00063 to 0.0008] | 0.00075 [0.0006 to 0.0008]
  Creatinine (g/dL)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Creatinine (g/dL)- Day42 | 0.00071 [0.00064 to 0.0008] | 0.0007 [0.00068 to 0.0008] | 0.0007 [0.00063 to 0.0008] | 0.00071 [0.0007 to 0.0008]
  Creatinine (g/dL)- Day98: number analyzed (Participants) | 32 | 36 | 0 | 21
  Creatinine (g/dL)- Day98 | 0.000705 [0.000615 to 0.00088] | 0.0008 [0.0007 to 0.00085] |  | 0.00072 [0.0007 to 0.0008]
  Creatinine (g/dL)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Creatinine (g/dL)- Day182 | 0.00073 [0.00064 to 0.0009] | 0.000715 [0.00068 to 0.0009] | 0.00078 [0.00067 to 0.00088] | 0.00077 [0.0007 to 0.0009]
  Creatinine (g/dL)- Day378: number analyzed (Participants) | 32 | 31 | 32 | 18
  Creatinine (g/dL)- Day378 | 0.00079 [0.0007 to 0.00088] | 0.00076 [0.0007 to 0.00084] | 0.0007 [0.000645 to 0.000835] | 0.0007 [0.00063 to 0.0008]
  Creatinine (g/dL)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Creatinine (g/dL)- Day455 | 0.000795 [0.00067 to 0.0009] | 0.00074 [0.0007 to 0.0009] | 0.00071 [0.000605 to 0.000835] | 0.0007 [0.00063 to 0.0009]

15. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin
Description: as for outcome 13
Time Frame: Measured during screening, Days 7, 42, 98, 182, 378, and 455
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
g/dL
  Hemoglobin (g/dL)- Screening | 13.75 [13.15 to 14.9] | 13.95 [12.9 to 15.2] | 13.85 [13.3 to 15.5] | 14.05 [13.25 to 14.9]
  Hemoglobin (g/dL)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Hemoglobin (g/dL)- Day7 | 13.5 [12.3 to 14.4] | 13.5 [12 to 14.3] | 13.4 [12.4 to 14.7] | 13.5 [12.4 to 14.5]
  Hemoglobin (g/dL)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Hemoglobin (g/dL)- Day42 | 13.7 [12.8 to 14.4] | 13.55 [12.8 to 14.5] | 13.65 [12.5 to 15] | 13.65 [12.9 to 14.7]
  Hemoglobin (g/dL)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Hemoglobin (g/dL)- Day98 | 13.35 [12.25 to 14.3] | 13.6 [12 to 14.3] |  | 13.2 [12.5 to 13.7]
  Hemoglobin (g/dL)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Hemoglobin (g/dL)- Day182 | 13.4 [12.4 to 14.1] | 13.5 [12.6 to 14.5] | 13.75 [12.2 to 14.9] | 13.25 [12.6 to 14.8]
  Hemoglobin (g/dL)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Hemoglobin (g/dL)- Day378 | 13.3 [12.45 to 14.05] | 13.5 [12 to 14] | 13.2 [11.8 to 14.4] | 13.3 [12.7 to 14]
  Hemoglobin (g/dL)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Hemoglobin (g/dL)- Day455 | 13.6 [12.6 to 14.3] | 13.8 [12.9 to 14.4] | 12.75 [12 to 14.6] | 13.6 [12.7 to 14.5]

16. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocytes, Neutrophils
Description: as for outcome 13
Time Frame: Measured during screening, Days 0, 1, 3, 7, 42, 84, 85, 87, 91, 98, 182, 378, and 455
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
thousand cells/cubic mm
  Lymphocytes (1000/cubic mm)- Screening | 2.1395 [1.7555 to 2.5785] | 2.095 [1.777 to 2.396] | 2.01 [1.6825 to 2.461] | 2.341 [2.0555 to 2.634]
  Lymphocytes (1000/cubic mm)- Day0: number analyzed (Participants) | 0 | 0 | 18 | 0
  Lymphocytes (1000/cubic mm)- Day0 |  |  | 2.0755 [1.66 to 2.283] |
  Lymphocytes (1000/cubic mm)- Day1: number analyzed (Participants) | 0 | 0 | 17 | 0
  Lymphocytes (1000/cubic mm)- Day1 |  |  | 1.982 [1.73 to 2.078] |
  Lymphocytes (1000/cubic mm)- Day3: number analyzed (Participants) | 0 | 0 | 15 | 0
  Lymphocytes (1000/cubic mm)- Day3 |  |  | 1.96 [1.547 to 2.166] |
  Lymphocytes (1000/cubic mm)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Lymphocytes (1000/cubic mm)- Day7 | 1.883 [1.6385 to 2.3735] | 1.93 [1.752 to 2.22] | 1.976 [1.622 to 2.445] | 2.2185 [1.738 to 2.571]
  Lymphocytes (1000/cubic mm)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Lymphocytes (1000/cubic mm)- Day42 | 1.76 [1.594 to 2.13] | 1.8915 [1.627 to 2.204] | 1.9915 [1.54 to 2.373] | 2.1375 [1.735 to 2.55]
  Lymphocytes (1000/cubic mm)- Day84: number analyzed (Participants) | 17 | 19 | 3 | 17
  Lymphocytes (1000/cubic mm)- Day84 | 1.891 [1.726 to 2.179] | 1.919 [1.624 to 2.29] | 1.99 [1.42 to 2.042] | 2.035 [1.75 to 2.298]
  Lymphocytes (1000/cubic mm)- Day85: number analyzed (Participants) | 16 | 16 | 0 | 13
  Lymphocytes (1000/cubic mm)- Day85 | 1.646 [1.327 to 2.119] | 1.7245 [1.4675 to 2.003] |  | 2.024 [1.763 to 2.589]
  Lymphocytes (1000/cubic mm)- Day87: number analyzed (Participants) | 18 | 13 | 0 | 13
  Lymphocytes (1000/cubic mm)- Day87 | 1.8725 [1.418 to 2.648] | 1.83 [1.659 to 2.157] |  | 2.076 [1.471 to 2.21]
  Lymphocytes (1000/cubic mm)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  Lymphocytes (1000/cubic mm)- Day91 | 1.8455 [1.522 to 2.302] | 2.02 [1.6795 to 2.36] |  | 2.036 [1.668 to 2.253]
  Lymphocytes (1000/cubic mm)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Lymphocytes (1000/cubic mm)- Day98 | 1.7605 [1.58 to 2.291] | 1.89 [1.601 to 2.247] |  | 2.085 [1.642 to 2.323]
  Lymphocytes (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Lymphocytes (1000/cubic mm)- Day182 | 1.969 [1.627 to 2.32] | 1.9905 [1.578 to 2.437] | 1.797 [1.481 to 2.17] | 1.9615 [1.751 to 2.263]
  Lymphocytes (1000/cubic mm)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Lymphocytes (1000/cubic mm)- Day378 | 1.7105 [1.487 to 2.102] | 1.859 [1.643 to 2.202] | 1.871 [1.543 to 2.211] | 2.0975 [1.608 to 2.321]
  Lymphocytes (1000/cubic mm)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Lymphocytes (1000/cubic mm)- Day455 | 1.753 [1.537 to 2.162] | 1.77 [1.51 to 2.087] | 1.9 [1.4515 to 2.1575] | 1.977 [1.548 to 2.22]
  Neutrophils (1000/cubic mm)- Screening | 2.9315 [2.29 to 5.254] | 2.9575 [2.154 to 4.3915] | 2.986 [1.88 to 3.7035] | 3.2245 [2.311 to 4.0635]
  Neutrophils (1000/cubic mm)- Day0: number analyzed (Participants) | 0 | 0 | 18 | 0
  Neutrophils (1000/cubic mm)- Day0 |  |  | 3.1935 [2.207 to 3.928] |
  Neutrophils (1000/cubic mm)- Day1: number analyzed (Participants) | 0 | 0 | 17 | 0
  Neutrophils (1000/cubic mm)- Day1 |  |  | 4.482 [3.854 to 5.877] |
  Neutrophils (1000/cubic mm)- Day3: number analyzed (Participants) | 0 | 0 | 15 | 0
  Neutrophils (1000/cubic mm)- Day3 |  |  | 2.82 [2.218 to 4.488] |
  Neutrophils (1000/cubic mm)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Neutrophils (1000/cubic mm)- Day7 | 2.903 [2.196 to 4.0295] | 2.84 [2.46 to 4.201] | 2.567 [1.9935 to 3.268] | 2.5425 [2.292 to 3.45]
  Neutrophils (1000/cubic mm)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Neutrophils (1000/cubic mm)- Day42 | 2.687 [1.863 to 3.2] | 2.9545 [2.246 to 3.605] | 2.6145 [1.761 to 3.142] | 2.679 [2.02 to 3.412]
  Neutrophils (1000/cubic mm)- Day84: number analyzed (Participants) | 17 | 19 | 3 | 17
  Neutrophils (1000/cubic mm)- Day84 | 3.065 [1.953 to 5.112] | 3.82 [2.521 to 4.914] | 1.739 [1.56 to 1.806] | 3.114 [2.024 to 3.748]
  Neutrophils (1000/cubic mm)- Day85: number analyzed (Participants) | 16 | 16 | 0 | 13
  Neutrophils (1000/cubic mm)- Day85 | 4.224 [3.41 to 5.2045] | 5.1475 [3.9985 to 6.6755] |  | 3.355 [2.415 to 3.872]
  Neutrophils (1000/cubic mm)- Day87: number analyzed (Participants) | 18 | 13 | 0 | 13
  Neutrophils (1000/cubic mm)- Day87 | 2.798 [1.794 to 4.522] | 3.214 [2.66 to 4.71] |  | 2.352 [1.868 to 3.389]
  Neutrophils (1000/cubic mm)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  Neutrophils (1000/cubic mm)- Day91 | 3.34 [2.42 to 4.598] | 3.65 [3.096 to 4.8395] |  | 3.407 [2.084 to 3.667]
  Neutrophils (1000/cubic mm)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Neutrophils (1000/cubic mm)- Day98 | 2.4375 [1.6465 to 3.898] | 2.814 [1.841 to 3.51] |  | 2.94 [2.157 to 3.657]
  Neutrophils (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Neutrophils (1000/cubic mm)- Day182 | 2.734 [1.83 to 3.304] | 2.4915 [1.811 to 3.812] | 2.3075 [1.78 to 2.844] | 2.6895 [2.324 to 3.412]
  Neutrophils (1000/cubic mm)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Neutrophils (1000/cubic mm)- Day378 | 2.6995 [2.0775 to 3.781] | 2.535 [1.92 to 3.34] | 2.292 [1.913 to 3.248] | 2.811 [2.13 to 3.41]
  Neutrophils (1000/cubic mm)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Neutrophils (1000/cubic mm)- Day455 | 2.5 [1.837 to 3.342] | 2.282 [1.748 to 3.921] | 2.2415 [1.77 to 3.1005] | 2.2905 [1.769 to 3.08]

17. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC
Description: as for outcome 13
Time Frame: Measured during screening, Days 0, 1, 3, 7, 42, 84, 85, 87, 91, 98, 182, 378, and 455
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
thousand cells/cubic mm
  WBC (1000/cubic mm)- Screening | 5.805 [5.015 to 8.18] | 5.5 [4.83 to 6.97] | 5.575 [4.23 to 6.57] | 6.415 [5.525 to 7.3]
  WBC (1000/cubic mm)- Day0: number analyzed (Participants) | 0 | 0 | 18 | 0
  WBC (1000/cubic mm)- Day0 |  |  | 5.67 [4.53 to 7.23] |
  WBC (1000/cubic mm)- Day1: number analyzed (Participants) | 0 | 0 | 17 | 0
  WBC (1000/cubic mm)- Day1 |  |  | 7.18 [6.49 to 8.53] |
  WBC (1000/cubic mm)- Day3: number analyzed (Participants) | 0 | 0 | 15 | 0
  WBC (1000/cubic mm)- Day3 |  |  | 5.74 [4.51 to 7.04] |
  WBC (1000/cubic mm)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  WBC (1000/cubic mm)- Day7 | 5.5 [4.49 to 7.07] | 5.56 [4.88 to 6.69] | 5.275 [4.24 to 6.005] | 5.36 [4.43 to 6.64]
  WBC (1000/cubic mm)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  WBC (1000/cubic mm)- Day42 | 4.89 [4.02 to 6.64] | 5.3 [4.63 to 6.09] | 5.05 [4.38 to 6.12] | 5.31 [4.09 to 6.17]
  WBC (1000/cubic mm)- Day84: number analyzed (Participants) | 17 | 19 | 3 | 17
  WBC (1000/cubic mm)- Day84 | 5.66 [4.19 to 7.33] | 5.95 [5.13 to 7.73] | 4.21 [3.86 to 4.48] | 5.42 [4.79 to 6.53]
  WBC (1000/cubic mm)- Day85: number analyzed (Participants) | 16 | 16 | 0 | 13
  WBC (1000/cubic mm)- Day85 | 6.965 [5.62 to 7.535] | 7.685 [6.38 to 9.15] |  | 5.8 [4.97 to 7.17]
  WBC (1000/cubic mm)- Day87: number analyzed (Participants) | 18 | 13 | 0 | 13
  WBC (1000/cubic mm)- Day87 | 5.55 [3.58 to 7.92] | 5.84 [5.31 to 7.38] |  | 4.88 [4.2 to 6.53]
  WBC (1000/cubic mm)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  WBC (1000/cubic mm)- Day91 | 6.39 [4.35 to 8.8] | 6.585 [5.275 to 7.03] |  | 5.305 [4.57 to 6.85]
  WBC (1000/cubic mm)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  WBC (1000/cubic mm)- Day98 | 4.935 [3.945 to 6.65] | 5.22 [4.54 to 6.18] |  | 5.5 [4.52 to 6.29]
  WBC (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  WBC (1000/cubic mm)- Day182 | 5.17 [4.22 to 6.61] | 5 [4.4 to 6.06] | 4.895 [4.19 to 5.98] | 5.405 [4.64 to 6.66]
  WBC (1000/cubic mm)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  WBC (1000/cubic mm)- Day378 | 5.37 [4.265 to 5.895] | 5.05 [4.07 to 5.75] | 5.06 [4.08 to 6.03] | 5.67 [4.62 to 6.06]
  WBC (1000/cubic mm)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  WBC (1000/cubic mm)- Day455 | 4.795 [3.55 to 6.61] | 4.62 [3.78 to 6.33] | 4.565 [4.035 to 5.675] | 4.745 [3.96 to 5.93]
  Platelets (1000/cubic mm)- Screening | 269.5 [232.5 to 321.5] | 269.5 [226.5 to 301.5] | 255.5 [224.5 to 298.5] | 260.5 [236 to 307]
  Platelets (1000/cubic mm)- Day0: number analyzed (Participants) | 0 | 0 | 18 | 0
  Platelets (1000/cubic mm)- Day0 |  |  | 269 [234 to 307] |
  Platelets (1000/cubic mm)- Day1: number analyzed (Participants) | 0 | 0 | 17 | 0
  Platelets (1000/cubic mm)- Day1 |  |  | 252 [232 to 292] |
  Platelets (1000/cubic mm)- Day3: number analyzed (Participants) | 0 | 0 | 15 | 0
  Platelets (1000/cubic mm)- Day3 |  |  | 242 [224 to 282] |
  Platelets (1000/cubic mm)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Platelets (1000/cubic mm)- Day7 | 269.5 [234.5 to 309] | 286 [232 to 305] | 256 [220 to 292] | 286 [239 to 306]
  Platelets (1000/cubic mm)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Platelets (1000/cubic mm)- Day42 | 267 [226 to 318] | 277 [238 to 307] | 256 [230 to 321] | 257.5 [244 to 302]
  Platelets (1000/cubic mm)- Day84: number analyzed (Participants) | 17 | 19 | 3 | 17
  Platelets (1000/cubic mm)- Day84 | 277 [251 to 311] | 261 [218 to 320] | 189 [126 to 250] | 271 [228 to 334]
  Platelets (1000/cubic mm)- Day85: number analyzed (Participants) | 16 | 16 | 0 | 13
  Platelets (1000/cubic mm)- Day85 | 272.5 [244 to 323.5] | 281 [237.5 to 318.5] |  | 272 [215 to 309]
  Platelets (1000/cubic mm)- Day87: number analyzed (Participants) | 18 | 13 | 0 | 13
  Platelets (1000/cubic mm)- Day87 | 283 [241 to 320] | 273 [237 to 319] |  | 265 [235 to 299]
  Platelets (1000/cubic mm)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  Platelets (1000/cubic mm)- Day91 | 286 [241 to 339] | 279.5 [256.5 to 309.5] |  | 289.5 [245 to 315]
  Platelets (1000/cubic mm)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Platelets (1000/cubic mm)- Day98 | 260 [235.5 to 317] | 256 [232 to 326] |  | 276 [231 to 321]
  Platelets (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Platelets (1000/cubic mm)- Day182 | 282 [239 to 306] | 272 [234 to 322] | 245.5 [222 to 287] | 256 [238 to 308]
  Platelets (1000/cubic mm)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Platelets (1000/cubic mm)- Day378 | 274 [243.5 to 316.5] | 282 [245 to 318] | 262 [241 to 314] | 275.5 [237 to 323]
  Platelets (1000/cubic mm)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Platelets (1000/cubic mm)- Day455 | 265.5 [220 to 308] | 275 [233 to 292] | 262 [219 to 292.5] | 259 [223 to 273]

18. Primary Outcome: Numbers of Participants With Grade 1 or Higher Local Laboratory Results
Description: The number (percentage) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the DAIDS AE Grading Table were tabulated by treatment arm for each post-vaccination time point.
Time Frame: Measured during screening, Days 0, 1, 3, 7, 42, 84, 85, 87, 91, 98, 182, 378, and 455
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  AST (U/L)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  AST (U/L)- Day7 | 0 | 0 | 0 | 1
  AST (U/L)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  AST (U/L)- Day42 | 1 | 1 | 0 | 2
  AST (U/L)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  AST (U/L)- Day98 | 1 | 1 |  | 0
  AST (U/L)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  AST (U/L)- Day182 | 0 | 0 | 2 | 0
  AST (U/L)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  AST (U/L)- Day378 | 0 | 0 | 2 | 1
  ALT (SGPT) (U/L)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  ALT (SGPT) (U/L)- Day7 | 0 | 1 | 0 | 0
  ALT (SGPT) (U/L)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  ALT (SGPT) (U/L)- Day42 | 2 | 1 | 1 | 1
  ALT (SGPT) (U/L)- Day84: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT (SGPT) (U/L)- Day84 |  |  | 1 |
  ALT (SGPT) (U/L)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  ALT (SGPT) (U/L)- Day98 | 1 | 1 |  | 0
  ALT (SGPT) (U/L)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  ALT (SGPT) (U/L)- Day182 | 0 | 0 | 1 | 0
  ALT (SGPT) (U/L)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  ALT (SGPT) (U/L)- Day378 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Hemoglobin (g/dL)- Day7 | 0 | 1 | 0 | 0
  Hemoglobin (g/dL)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Hemoglobin (g/dL)- Day42 | 1 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day84: number analyzed (Participants) | 17 | 19 | 3 | 17
  Hemoglobin (g/dL)- Day84 | 0 | 0 | 0 | 2
  Hemoglobin (g/dL)- Day85: number analyzed (Participants) | 16 | 16 | 0 | 13
  Hemoglobin (g/dL)- Day85 | 0 | 1 |  | 0
  Hemoglobin (g/dL)- Day87: number analyzed (Participants) | 18 | 13 | 0 | 13
  Hemoglobin (g/dL)- Day87 | 0 | 1 |  | 0
  Hemoglobin (g/dL)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  Hemoglobin (g/dL)- Day91 | 0 | 1 |  | 1
  Hemoglobin (g/dL)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Hemoglobin (g/dL)- Day98 | 0 | 1 |  | 1
  Hemoglobin (g/dL)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Hemoglobin (g/dL)- Day182 | 0 | 2 | 1 | 0
  Hemoglobin (g/dL)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Hemoglobin (g/dL)- Day378 | 2 | 2 | 0 | 0
  Hemoglobin (g/dL)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Hemoglobin (g/dL)- Day455 | 0 | 1 | 0 | 0
  Creatinine (g/dL)- Day7: number analyzed (Participants) | 36 | 33 | 33 | 22
  Creatinine (g/dL)- Day7 | 4 | 1 | 1 | 2
  Creatinine (g/dL)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Creatinine (g/dL)- Day42 | 3 | 1 | 0 | 0
  Creatinine (g/dL)- Day84: number analyzed (Participants) | 3 | 0 | 0 | 0
  Creatinine (g/dL)- Day84 | 1 |  |  |
  Creatinine (g/dL)- Day98: number analyzed (Participants) | 32 | 36 | 0 | 21
  Creatinine (g/dL)- Day98 | 4 | 4 |  | 0
  Creatinine (g/dL)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Creatinine (g/dL)- Day182 | 3 | 2 | 3 | 0
  Creatinine (g/dL)- Day378: number analyzed (Participants) | 32 | 31 | 32 | 18
  Creatinine (g/dL)- Day378 | 4 | 1 | 1 | 0
  Creatinine (g/dL)- Day455: number analyzed (Participants) | 30 | 31 | 32 | 18
  Creatinine (g/dL)- Day455 | 1 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day7: number analyzed (Participants) | 36 | 33 | 32 | 22
  Platelets (1000/cubic mm)- Day7 | 0 | 0 | 1 | 0
  Platelets (1000/cubic mm)- Day42: number analyzed (Participants) | 33 | 34 | 34 | 22
  Platelets (1000/cubic mm)- Day42 | 0 | 0 | 1 | 0
  Platelets (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Platelets (1000/cubic mm)- Day182 | 0 | 0 | 1 | 0
  Neutrophils (1000/cubic mm)- Day91: number analyzed (Participants) | 18 | 16 | 0 | 14
  Neutrophils (1000/cubic mm)- Day91 | 1 | 0 |  | 0
  Neutrophils (1000/cubic mm)- Day98: number analyzed (Participants) | 32 | 35 | 0 | 21
  Neutrophils (1000/cubic mm)- Day98 | 1 | 0 |  | 0
  Neutrophils (1000/cubic mm)- Day182: number analyzed (Participants) | 31 | 30 | 34 | 18
  Neutrophils (1000/cubic mm)- Day182 | 1 | 1 | 0 | 0
  Neutrophils (1000/cubic mm)- Day378: number analyzed (Participants) | 32 | 31 | 31 | 18
  Neutrophils (1000/cubic mm)- Day378 | 1 | 1 | 1 | 0

19. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: There were no early study terminations associated with an AE or reactogenicity reported by any participant.
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) gp120/MF59 mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120/MF59® (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
- Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) gp120+Alum mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120 (an admixture of 100 mcg of TV1.C gp120 and 100 mcg of 1806.C gp120) admixed with Aluminum Hydroxide Suspension to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
- Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12)p120/MF59 mo(0,1,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 6, and 12 AND Bivalent Subtype C gp120/MF59® (an admixture of 100 mcg of TV1.C gp120, 100 mcg of 1086.C gp120, and MF59C.1) to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 0, 1, 6, and 12
- Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12) gp120 mo(3,6,12): ALVAC-HIV (vCP2438) to be administered as 1 mL IM in LEFT deltoid (unless medically contraindicated) at months 0, 1, 3, 6, and 12 AND Bivalent Subtype C gp120 (an admixture of 100 mcg of TV1.C gp120 and 100 mcg of 1806.C gp120) admixed with Sodium Chloride for Injection, 0.9% to be administered as 0.5mL IM in RIGHT deltoid (unless medically contraindicated) at Months 3, 6, and 12
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12)p120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12) gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product discontinuation reasons are tabulated by treatment arm.
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 36 | 36 | 36 | 24
Participants
  Clinical event other than reactogenicity | 1 | 1 | 0 | 0
  Reactogenicity | 0 | 0 | 0 | 0
  Other reason | 4 | 3 | 4 | 6
  No discontinuation | 31 | 32 | 32 | 18

21. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C)
Description: as for outcome 1
Time Frame: Measured at Months 6.5 and 12.
Population: Overall Number of Participants Analyzed represents the number of enrolled participants with available specimens. "Number Analyzed" shows the number of HIV uninfected participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 29 | 28 | 33 | 17
Participants
  1086C_D7gp120.avi/293F (Month 6.5): number analyzed (Participants) | 29 | 27 | 33 | 17
  1086C_D7gp120.avi/293F (Month 6.5) | 29 | 26 | 32 | 17
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 28 | 28 | 32 | 17
  96ZM651.D11gp120.avi (Month 6.5) | 27 | 27 | 30 | 17
  TV1c8_D11gp120.avi/293F (Month 6.5) | 29 | 27 | 32 | 17
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 29 | 27 | 31 | 17
  1086C_D7gp120.avi/293F (Month 12) | 29 | 26 | 29 | 17
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 28 | 28 | 29 | 16
  96ZM651.D11gp120.avi (Month 12) | 7 | 5 | 25 | 1
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  TV1c8_D11gp120.avi/293F (Month 12) | 25 | 22 | 29 | 12

22. Secondary Outcome: Level of Vaccine-induced Serum IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C)
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Summary was calculated among positive responders only (positivity criteria are described in Outcome 1).
Time Frame: Measured at Months 6.5 and 12.
Population: "Overall Number of Participants Analyzed" represents the number of enrolled participants with available specimens. "Number Analyzed" shows the number of HIV uninfected participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 28 | 32 | 17
relative fluorescence units
  1086C_D7gp120.avi/293F (Month 6.5): number analyzed (Participants) | 29 | 26 | 32 | 17
  1086C_D7gp120.avi/293F (Month 6.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 27 | 27 | 30 | 17
  96ZM651.D11gp120.avi (Month 6.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [13363 to 22000]
  TV1c8_D11gp120.avi/293F (Month 6.5): number analyzed (Participants) | 29 | 27 | 32 | 17
  TV1c8_D11gp120.avi/293F (Month 6.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 29 | 26 | 29 | 17
  1086C_D7gp120.avi/293F (Month 12) | 6759.8 [3662.2 to 15765.5] | 11657.1 [3131.1 to 18042.6] | 22000 [13782 to 22000] | 4265.8 [2385 to 8666.5]
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 7 | 5 | 25 | 1
  96ZM651.D11gp120.avi (Month 12) | 3182.8 [1705.4 to 4285.9] | 2167.8 [1767.5 to 2524.8] | 3000 [1871.5 to 6561] | 1676 [1676 to 1676]
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 25 | 22 | 29 | 12
  TV1c8_D11gp120.avi/293F (Month 12) | 1252.5 [686 to 3761.2] | 1660 [892.6 to 2898.4] | 10750 [5326.5 to 22000] | 1086 [442.6 to 2429.1]
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 30 | 27 | 31 | 16
  1086C_D7gp120.avi/293F (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 26 | 28 | 30 | 15
  96ZM651.D11gp120.avi (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 28 | 28 | 29 | 15
  TV1c8_D11gp120.avi/293F (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 27 | 27 | 32 | 16
  1086C_D7gp120.avi/293F (Month 18) | 22000 [13447.4 to 22000] | 22000 [17031.4 to 22000] | 22000 [16465.8 to 22000] | 16187 [8260.8 to 22000]
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 17 | 22 | 28 | 7
  96ZM651.D11gp120.avi (Month 18) | 6135.8 [4058.2 to 10887] | 5439 [2617.8 to 8736.1] | 5372.6 [3140.4 to 12123.9] | 2794 [2226 to 4364.1]
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 26 | 28 | 30 | 15
  TV1c8_D11gp120.avi/293F (Month 18) | 8367.6 [2745.8 to 21097.6] | 8893.4 [3450.6 to 20507.7] | 20549 [8176.7 to 22000] | 6794.5 [2788.2 to 9961.5]

23. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG Ab Binding to V2 Env Proteins
Description: as for outcome 1
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 29 | 28 | 33 | 17
Participants
  00MSA 4076 gp140 (Month 6.5) | 27 | 27 | 30 | 15
  A1.con.env03 140 CF (Month 6.5) | 27 | 27 | 31 | 17
  AE.A244 V1V2 Tags/293F (Month 6.5) | 22 | 23 | 28 | 11
  C.1086C_V1_V2 Tags (Month 6.5) | 14 | 13 | 16 | 2
  Con 6 gp120/B (Month 6.5) | 26 | 26 | 29 | 17
  Con S gp140 CFI (Month 6.5) | 29 | 27 | 32 | 17
  gp41 (Month 6.5): number analyzed (Participants) | 29 | 27 | 32 | 17
  gp41 (Month 6.5) | 0 | 1 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 6.5): number analyzed (Participants) | 24 | 27 | 29 | 16
  gp70-96ZM651.02 V1v2 (Month 6.5) | 8 | 13 | 19 | 4
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 26 | 27 | 30 | 17
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 17 | 15 | 26 | 4
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 27 | 27 | 30 | 17
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 10 | 14 | 24 | 4
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 26 | 27 | 30 | 17
  gp70_B.CaseA_V1_V2 (Month 6.5) | 9 | 13 | 25 | 3
  00MSA 4076 gp140 (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  00MSA 4076 gp140 (Month 12) | 4 | 1 | 12 | 1
  A1.con.env03 140 CF (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  A1.con.env03 140 CF (Month 12) | 15 | 14 | 25 | 5
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  AE.A244 V1V2 Tags/293F (Month 12) | 4 | 6 | 6 | 1
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  C.1086C_V1_V2 Tags (Month 12) | 0 | 0 | 0 | 1
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 16
  Con 6 gp120/B (Month 12) | 3 | 1 | 14 | 1
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 29 | 28 | 31 | 17
  Con S gp140 CFI (Month 12) | 22 | 25 | 30 | 13
  gp41 (Month 12): number analyzed (Participants) | 29 | 27 | 30 | 17
  gp41 (Month 12) | 0 | 0 | 0 | 1
  gp70-96ZM651.02 V1v2 (Month 12): number analyzed (Participants) | 25 | 27 | 27 | 15
  gp70-96ZM651.02 V1v2 (Month 12) | 0 | 1 | 2 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 26 | 27 | 28 | 16
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 1 | 2 | 6 | 1
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 27 | 27 | 28 | 16
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 1 | 2 | 3 | 0
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 26 | 27 | 28 | 16
  gp70_B.CaseA_V1_V2 (Month 12) | 1 | 1 | 4 | 0

24. Secondary Outcome: Level of Vaccine-induced Serum IgG Ab Binding to V2 Env Proteins
Description: as for outcome 22
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 28 | 32 | 17
relative fluorescence units
  00MSA 4076 gp140 (Month 6.5): number analyzed (Participants) | 27 | 27 | 30 | 15
  00MSA 4076 gp140 (Month 6.5) | 18852.2 [10385.8 to 22000] | 11851.2 [4795.8 to 20954.4] | 22000 [19705.7 to 22000] | 9648.8 [4793.4 to 18959]
  A1.con.env03 140 CF (Month 6.5): number analyzed (Participants) | 27 | 27 | 31 | 17
  A1.con.env03 140 CF (Month 6.5) | 21481.5 [10941 to 22000] | 15307.5 [7928.9 to 22000] | 22000 [19518.4 to 22000] | 12791.2 [6158.2 to 21474]
  AE.A244 V1V2 Tags/293F (Month 6.5): number analyzed (Participants) | 22 | 23 | 28 | 11
  AE.A244 V1V2 Tags/293F (Month 6.5) | 7008.2 [1079.8 to 9841.2] | 4347.5 [2171.8 to 7081.4] | 3203 [1343.1 to 10818.8] | 489 [409.5 to 2427.8]
  C.1086C_V1_V2 Tags (Month 6.5): number analyzed (Participants) | 14 | 13 | 16 | 2
  C.1086C_V1_V2 Tags (Month 6.5) | 1284.5 [1139.7 to 1831.6] | 954.5 [866.2 to 3260] | 1830.8 [1104.4 to 2254.2] | 865.6 [796.6 to 934.7]
  Con 6 gp120/B (Month 6.5): number analyzed (Participants) | 26 | 26 | 29 | 17
  Con 6 gp120/B (Month 6.5) | 21899.6 [11363.6 to 22000] | 14046.6 [9418.1 to 22000] | 22000 [22000 to 22000] | 9978 [5492 to 20428.5]
  Con S gp140 CFI (Month 6.5): number analyzed (Participants) | 29 | 27 | 32 | 17
  Con S gp140 CFI (Month 6.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  gp41 (Month 6.5): number analyzed (Participants) | 0 | 1 | 0 | 0
  gp41 (Month 6.5) |  | 4472.8 [4472.8 to 4472.8] |  |
  gp70-96ZM651.02 V1v2 (Month 6.5): number analyzed (Participants) | 8 | 13 | 19 | 4
  gp70-96ZM651.02 V1v2 (Month 6.5) | 968 [745.2 to 1412.3] | 1963 [1040.5 to 4739.8] | 2631.8 [1444 to 6033.8] | 1219.4 [695.3 to 1835.2]
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 17 | 15 | 26 | 4
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 714.8 [386.5 to 1925] | 1367.5 [916.9 to 4679.8] | 6205.1 [1550.6 to 13995.4] | 727.1 [430.1 to 1152.1]
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 10 | 14 | 24 | 4
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 1476 [587.5 to 3383] | 1888.8 [1204.9 to 4129] | 6450.5 [1593.2 to 8631.6] | 406.9 [355.6 to 725.1]
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 9 | 13 | 25 | 3
  gp70_B.CaseA_V1_V2 (Month 6.5) | 1368.8 [727 to 3992.5] | 1292.5 [819.5 to 5713.8] | 4521.2 [1193.5 to 10484] | 651.8 [520.8 to 1328.8]
  00MSA 4076 gp140 (Month 12): number analyzed (Participants) | 4 | 1 | 12 | 1
  00MSA 4076 gp140 (Month 12) | 1557.1 [919.9 to 2207.1] | 1390.2 [1390.2 to 1390.2] | 1425.8 [1151.9 to 2257.9] | 952 [952 to 952]
  A1.con.env03 140 CF (Month 12): number analyzed (Participants) | 15 | 14 | 25 | 5
  A1.con.env03 140 CF (Month 12) | 286.5 [199.6 to 483.8] | 318.1 [206.5 to 527.6] | 834.8 [360 to 1718] | 339.2 [169.8 to 709.2]
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 4 | 6 | 6 | 1
  AE.A244 V1V2 Tags/293F (Month 12) | 290.4 [226 to 497.6] | 237.5 [196.7 to 270.4] | 279.2 [245.8 to 309.8] | 124.2 [124.2 to 124.2]
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 1
  C.1086C_V1_V2 Tags (Month 12) |  |  |  | 1296.8 [1296.8 to 1296.8]
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 3 | 1 | 14 | 1
  Con 6 gp120/B (Month 12) | 2429.8 [1981.9 to 3020.2] | 1139.8 [1139.8 to 1139.8] | 1908.5 [1479.8 to 2280.8] | 2036.8 [2036.8 to 2036.8]
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 22 | 25 | 30 | 13
  Con S gp140 CFI (Month 12) | 954 [556.6 to 2888.4] | 1599 [916.2 to 2333.5] | 6908.8 [2639.8 to 14532.9] | 680.2 [397 to 1169]
  gp41 (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 1
  gp41 (Month 12) |  |  |  | 9264 [9264 to 9264]
  gp70-96ZM651.02 V1v2 (Month 12): number analyzed (Participants) | 0 | 1 | 2 | 0
  gp70-96ZM651.02 V1v2 (Month 12) |  | 1264.8 [1264.8 to 1264.8] | 819.9 [561.7 to 1078.1] |
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 1 | 2 | 6 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 495.2 [495.2 to 495.2] | 502.4 [421.6 to 583.2] | 722.4 [218.6 to 1481.9] | 2504.8 [2504.8 to 2504.8]
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 1 | 2 | 3 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 693.8 [693.8 to 693.8] | 559.9 [490.7 to 629.1] | 427 [378.2 to 1999.4] |
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 1 | 1 | 4 | 0
  gp70_B.CaseA_V1_V2 (Month 12) | 949 [949 to 949] | 442.5 [442.5 to 442.5] | 487.2 [283.1 to 1070] |
  00MSA 4076 gp140 (Month 12.5): number analyzed (Participants) | 26 | 28 | 29 | 15
  00MSA 4076 gp140 (Month 12.5) | 22000 [18877.6 to 22000] | 22000 [13449.4 to 22000] | 22000 [17787.8 to 22000] | 22000 [11267.2 to 22000]
  A1.con.env03 140 CF (Month 12.5): number analyzed (Participants) | 27 | 28 | 29 | 15
  A1.con.env03 140 CF (Month 12.5) | 22000 [20752 to 22000] | 22000 [17453.4 to 22000] | 22000 [22000 to 22000] | 22000 [16264.4 to 22000]
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 21 | 27 | 27 | 14
  AE.A244 V1V2 Tags/293F (Month 12.5) | 4553.5 [2286.2 to 9393.8] | 3313.8 [1245.9 to 10641.6] | 5728.8 [2011.8 to 10929.1] | 1034.2 [482.6 to 5401.9]
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 19 | 21 | 22 | 9
  C.1086C_V1_V2 Tags (Month 12.5) | 2021.2 [1142.2 to 3862.8] | 3476 [906 to 6288.5] | 3484.6 [994 to 8674.6] | 1380.2 [601 to 3883]
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 26 | 28 | 29 | 15
  Con 6 gp120/B (Month 12.5) | 22000 [22000 to 22000] | 22000 [20433.4 to 22000] | 22000 [22000 to 22000] | 22000 [15222.2 to 22000]
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 28 | 28 | 30 | 15
  Con S gp140 CFI (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  gp41 (Month 12.5): number analyzed (Participants) | 0 | 0 | 3 | 2
  gp41 (Month 12.5) |  |  | 4644.8 [3651.8 to 13322.4] | 8348.5 [5951.1 to 10745.9]
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 10 | 18 | 18 | 7
  gp70-96ZM651.02 V1v2 (Month 12.5) | 1427.2 [891.8 to 9947.6] | 3770.8 [1125 to 10077.4] | 8793.6 [1318.6 to 21615.9] | 1639.8 [1290.2 to 6055.9]
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 16 | 25 | 24 | 9
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 1407.4 [993.3 to 3027.4] | 2057.8 [714.5 to 6260.2] | 12436.5 [1806.4 to 22000] | 2031.8 [1158.8 to 4055.5]
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 12 | 22 | 23 | 8
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 1213.2 [734.6 to 3588.6] | 2332.9 [732.9 to 5249.1] | 8987.2 [2613.6 to 22000] | 1324.4 [941.3 to 3481.6]
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 11 | 20 | 22 | 6
  gp70_B.CaseA_V1_V2 (Month 12.5) | 763.5 [670.1 to 3615.2] | 2246.5 [999.1 to 5417.9] | 8372.5 [1587.8 to 21441.9] | 2869.5 [1171.8 to 4368.3]
  00MSA 4076 gp140 (Month 18): number analyzed (Participants) | 11 | 12 | 18 | 4
  00MSA 4076 gp140 (Month 18) | 1954 [1242.2 to 3022] | 2546.9 [1072.2 to 7260.1] | 1571 [1131.2 to 3575.8] | 1351.9 [1189.6 to 1367.8]
  A1.con.env03 140 CF (Month 18): number analyzed (Participants) | 23 | 26 | 29 | 11
  A1.con.env03 140 CF (Month 18) | 1106 [444.2 to 2628] | 1552.5 [607 to 3231.8] | 1853.2 [929.5 to 4194.5] | 961.5 [695.8 to 1429.6]
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 5 | 9 | 12 | 2
  AE.A244 V1V2 Tags/293F (Month 18) | 137 [110.2 to 484] | 462 [371.2 to 512.5] | 362.2 [194.8 to 1003.6] | 445.9 [429.3 to 462.4]
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 1 | 3 | 3 | 1
  C.1086C_V1_V2 Tags (Month 18) | 1204.5 [1204.5 to 1204.5] | 1523.2 [1067.4 to 5288.9] | 821.8 [714.1 to 2419.4] | 909 [909 to 909]
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 13 | 17 | 25 | 6
  Con 6 gp120/B (Month 18) | 2373.2 [1574 to 4438.2] | 2805 [1459.5 to 4348.8] | 2405.5 [1517.5 to 4459.5] | 1185.2 [993.6 to 1463.2]
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 25 | 28 | 31 | 15
  Con S gp140 CFI (Month 18) | 8793.8 [3178.8 to 16947.8] | 9031.1 [3772.2 to 22000] | 13261.8 [7458.2 to 22000] | 5032.5 [3082 to 9318.4]
  gp41 (Month 18): number analyzed (Participants) | 0 | 1 | 3 | 1
  gp41 (Month 18) |  | 2549.2 [2549.2 to 2549.2] | 7284.8 [5785.5 to 14642.4] | 19096.5 [19096.5 to 19096.5]
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 1 | 3 | 4 | 1
  gp70-96ZM651.02 V1v2 (Month 18) | 370.8 [370.8 to 370.8] | 584 [541.4 to 872.1] | 987.8 [590.4 to 1672.9] | 2221.8 [2221.8 to 2221.8]
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 4 | 10 | 11 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 163.1 [125.2 to 272.5] | 180.2 [130.4 to 208.4] | 1319.2 [605.5 to 1729.8] | 1114.2 [1114.2 to 1114.2]
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 1 | 3 | 7 | 1
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 244.5 [244.5 to 244.5] | 1593.8 [914.8 to 1638.4] | 1332 [425 to 1556] | 1227.5 [1227.5 to 1227.5]
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 1 | 2 | 6 | 1
  gp70_B.CaseA_V1_V2 (Month 18) | 314.2 [314.2 to 314.2] | 1717.6 [1210.9 to 2224.3] | 623.8 [383.3 to 886.9] | 593.2 [593.2 to 593.2]

25. Secondary Outcome: Vaccine-induced Occurrence of CD4+ T-cells Expressing Markers in Response to HIV Proteins Included in the Vaccine
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers (IFNg and/or IL-2) after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if adjusted p-value <=0.00001. Any Env magnitude is the maximum of 1086 gp120, TV1 gp120, and Env ZM96 magnitudes. Any HIV magnitude is the sum of Any Env and LAI Gag magnitudes. Data are excluded if blood draw date was outside the visit window, participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at Months 6.5, 12, 12.5, and 18
Population: "Overall Number of Participants Analyzed" represents the number of enrolled participants with available specimens. "Number Analyzed" shows the number of HIV uninfected participants with available ICS data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 32 | 31 | 32 | 18
Participants
  1086 gp120 (Month 6.5): number analyzed (Participants) | 31 | 29 | 31 | 18
  1086 gp120 (Month 6.5) | 15 | 19 | 16 | 6
  Any Env (Month 6.5): number analyzed (Participants) | 23 | 26 | 26 | 18
  Any Env (Month 6.5) | 16 | 20 | 21 | 8
  Any HIV (Month 6.5): number analyzed (Participants) | 23 | 26 | 26 | 18
  Any HIV (Month 6.5) | 17 | 20 | 21 | 8
  Env ZM96 (Month 6.5): number analyzed (Participants) | 23 | 26 | 26 | 18
  Env ZM96 (Month 6.5) | 12 | 14 | 8 | 5
  Env-1-ZM96 (Month 6.5): number analyzed (Participants) | 31 | 29 | 31 | 18
  Env-1-ZM96 (Month 6.5) | 12 | 15 | 7 | 5
  Env-2-ZM96 (Month 6.5): number analyzed (Participants) | 31 | 29 | 31 | 18
  Env-2-ZM96 (Month 6.5) | 3 | 5 | 6 | 1
  LAI Gag (Month 6.5): number analyzed (Participants) | 31 | 29 | 31 | 18
  LAI Gag (Month 6.5) | 1 | 0 | 1 | 2
  TV1 gp120 (Month 6.5): number analyzed (Participants) | 31 | 29 | 31 | 18
  TV1 gp120 (Month 6.5) | 15 | 20 | 20 | 6
  1086 gp120 (Month 12): number analyzed (Participants) | 30 | 30 | 30 | 17
  1086 gp120 (Month 12) | 6 | 13 | 10 | 0
  Any Env (Month 12): number analyzed (Participants) | 27 | 28 | 28 | 16
  Any Env (Month 12) | 9 | 16 | 13 | 5
  Any HIV (Month 12): number analyzed (Participants) | 27 | 28 | 28 | 16
  Any HIV (Month 12) | 10 | 16 | 14 | 5
  Env ZM96 (Month 12): number analyzed (Participants) | 27 | 28 | 28 | 16
  Env ZM96 (Month 12) | 6 | 9 | 4 | 4
  Env-1-ZM96 (Month 12): number analyzed (Participants) | 30 | 30 | 31 | 17
  Env-1-ZM96 (Month 12) | 6 | 9 | 4 | 5
  Env-2-ZM96 (Month 12): number analyzed (Participants) | 30 | 30 | 31 | 17
  Env-2-ZM96 (Month 12) | 1 | 4 | 2 | 0
  LAI Gag (Month 12): number analyzed (Participants) | 30 | 30 | 31 | 17
  LAI Gag (Month 12) | 1 | 2 | 1 | 1
  TV1 gp120 (Month 12): number analyzed (Participants) | 30 | 30 | 31 | 17
  TV1 gp120 (Month 12) | 8 | 17 | 13 | 2
  1086 gp120 (Month 12.5): number analyzed (Participants) | 32 | 31 | 31 | 17
  1086 gp120 (Month 12.5) | 15 | 21 | 12 | 5
  Any Env (Month 12.5): number analyzed (Participants) | 30 | 30 | 29 | 15
  Any Env (Month 12.5) | 25 | 24 | 18 | 9
  Any HIV (Month 12.5): number analyzed (Participants) | 30 | 30 | 29 | 15
  Any HIV (Month 12.5) | 25 | 24 | 19 | 9
  Env ZM96 (Month 12.5): number analyzed (Participants) | 30 | 30 | 29 | 15
  Env ZM96 (Month 12.5) | 15 | 20 | 6 | 8
  Env-1-ZM96 (Month 12.5): number analyzed (Participants) | 32 | 31 | 31 | 17
  Env-1-ZM96 (Month 12.5) | 15 | 20 | 5 | 9
  Env-2-ZM96 (Month 12.5): number analyzed (Participants) | 32 | 31 | 31 | 17
  Env-2-ZM96 (Month 12.5) | 1 | 8 | 4 | 0
  LAI Gag (Month 12.5): number analyzed (Participants) | 32 | 31 | 31 | 17
  LAI Gag (Month 12.5) | 1 | 2 | 1 | 1
  TV1 gp120 (Month 12.5): number analyzed (Participants) | 32 | 31 | 31 | 17
  TV1 gp120 (Month 12.5) | 20 | 24 | 16 | 8
  1086 gp120 (Month 18): number analyzed (Participants) | 29 | 31 | 32 | 16
  1086 gp120 (Month 18) | 9 | 21 | 10 | 5
  Any Env (Month 18): number analyzed (Participants) | 28 | 29 | 31 | 16
  Any Env (Month 18) | 16 | 23 | 13 | 9
  Any HIV (Month 18): number analyzed (Participants) | 28 | 29 | 31 | 16
  Any HIV (Month 18) | 17 | 23 | 14 | 9
  Env ZM96 (Month 18): number analyzed (Participants) | 28 | 29 | 31 | 16
  Env ZM96 (Month 18) | 14 | 18 | 4 | 6
  Env-1-ZM96 (Month 18): number analyzed (Participants) | 29 | 31 | 32 | 16
  Env-1-ZM96 (Month 18) | 14 | 20 | 3 | 6
  Env-2-ZM96 (Month 18): number analyzed (Participants) | 29 | 31 | 32 | 16
  Env-2-ZM96 (Month 18) | 0 | 4 | 2 | 0
  LAI Gag (Month 18): number analyzed (Participants) | 29 | 31 | 32 | 16
  LAI Gag (Month 18) | 1 | 2 | 1 | 0
  TV1 gp120 (Month 18): number analyzed (Participants) | 29 | 31 | 32 | 16
  TV1 gp120 (Month 18) | 11 | 23 | 11 | 7

26. Secondary Outcome: Vaccine-induced Percentage of CD4+ T-cells Expressing Markers in Response to HIV Proteins Included in the Vaccine
Description: as for outcome 25
Time Frame: Measured at Months 6.5, 12, 12.5, and 18
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 25 | 24 | 21 | 9
% CD4+ T-cells
  1086 gp120 (Month 6.5): number analyzed (Participants) | 15 | 19 | 16 | 6
  1086 gp120 (Month 6.5) | 0.209 [0.115 to 0.259] | 0.181 [0.123 to 0.277] | 0.222 [0.08 to 0.294] | 0.124 [0.108 to 0.161]
  Any Env (Month 6.5): number analyzed (Participants) | 16 | 20 | 21 | 8
  Any Env (Month 6.5) | 0.216 [0.136 to 0.339] | 0.182 [0.145 to 0.407] | 0.149 [0.121 to 0.332] | 0.142 [0.115 to 0.209]
  Any HIV (Month 6.5): number analyzed (Participants) | 17 | 20 | 21 | 8
  Any HIV (Month 6.5) | 0.221 [0.136 to 0.358] | 0.221 [0.158 to 0.43] | 0.202 [0.118 to 0.319] | 0.148 [0.135 to 0.291]
  Env ZM96 (Month 6.5): number analyzed (Participants) | 12 | 14 | 8 | 5
  Env ZM96 (Month 6.5) | 0.224 [0.104 to 0.339] | 0.162 [0.142 to 0.276] | 0.237 [0.194 to 0.255] | 0.137 [0.133 to 0.262]
  Env-1-ZM96 (Month 6.5): number analyzed (Participants) | 12 | 15 | 7 | 5
  Env-1-ZM96 (Month 6.5) | 0.186 [0.078 to 0.269] | 0.151 [0.098 to 0.233] | 0.16 [0.136 to 0.162] | 0.13 [0.117 to 0.189]
  Env-2-ZM96 (Month 6.5): number analyzed (Participants) | 3 | 5 | 6 | 1
  Env-2-ZM96 (Month 6.5) | 0.107 [0.1 to 0.147] | 0.067 [0.059 to 0.102] | 0.097 [0.084 to 0.111] | 0.072 [0.072 to 0.072]
  LAI Gag (Month 6.5): number analyzed (Participants) | 1 | 0 | 1 | 2
  LAI Gag (Month 6.5) | 0.108 [0.108 to 0.108] |  | 0.09 [0.09 to 0.09] | 0.092 [0.082 to 0.102]
  TV1 gp120 (Month 6.5): number analyzed (Participants) | 15 | 20 | 20 | 6
  TV1 gp120 (Month 6.5) | 0.193 [0.114 to 0.258] | 0.175 [0.135 to 0.326] | 0.152 [0.11 to 0.275] | 0.132 [0.104 to 0.184]
  1086 gp120 (Month 12): number analyzed (Participants) | 6 | 13 | 10 | 0
  1086 gp120 (Month 12) | 0.173 [0.156 to 0.199] | 0.157 [0.117 to 0.322] | 0.153 [0.127 to 0.177] |
  Any Env (Month 12): number analyzed (Participants) | 9 | 16 | 13 | 5
  Any Env (Month 12) | 0.15 [0.119 to 0.286] | 0.185 [0.116 to 0.298] | 0.156 [0.095 to 0.255] | 0.124 [0.089 to 0.176]
  Any HIV (Month 12): number analyzed (Participants) | 10 | 16 | 14 | 5
  Any HIV (Month 12) | 0.149 [0.104 to 0.281] | 0.206 [0.134 to 0.317] | 0.161 [0.11 to 0.264] | 0.167 [0.124 to 0.172]
  Env ZM96 (Month 12): number analyzed (Participants) | 6 | 9 | 4 | 4
  Env ZM96 (Month 12) | 0.238 [0.131 to 0.307] | 0.146 [0.13 to 0.365] | 0.157 [0.133 to 0.197] | 0.133 [0.083 to 0.178]
  Env-1-ZM96 (Month 12): number analyzed (Participants) | 6 | 9 | 4 | 5
  Env-1-ZM96 (Month 12) | 0.215 [0.134 to 0.225] | 0.125 [0.092 to 0.196] | 0.085 [0.077 to 0.128] | 0.107 [0.089 to 0.17]
  Env-2-ZM96 (Month 12): number analyzed (Participants) | 1 | 4 | 2 | 0
  Env-2-ZM96 (Month 12) | 0.101 [0.101 to 0.101] | 0.113 [0.056 to 0.172] | 0.072 [0.066 to 0.077] |
  LAI Gag (Month 12): number analyzed (Participants) | 1 | 2 | 1 | 1
  LAI Gag (Month 12) | 0.065 [0.065 to 0.065] | 0.053 [0.05 to 0.056] | 0.159 [0.159 to 0.159] | 0.056 [0.056 to 0.056]
  TV1 gp120 (Month 12): number analyzed (Participants) | 8 | 17 | 13 | 2
  TV1 gp120 (Month 12) | 0.124 [0.095 to 0.286] | 0.172 [0.109 to 0.237] | 0.118 [0.089 to 0.219] | 0.087 [0.078 to 0.097]
  1086 gp120 (Month 12.5): number analyzed (Participants) | 15 | 21 | 12 | 5
  1086 gp120 (Month 12.5) | 0.118 [0.097 to 0.189] | 0.158 [0.13 to 0.298] | 0.142 [0.104 to 0.259] | 0.161 [0.105 to 0.18]
  Any Env (Month 12.5): number analyzed (Participants) | 25 | 24 | 18 | 9
  Any Env (Month 12.5) | 0.172 [0.105 to 0.215] | 0.277 [0.148 to 0.472] | 0.138 [0.103 to 0.236] | 0.18 [0.096 to 0.207]
  Any HIV (Month 12.5): number analyzed (Participants) | 25 | 24 | 19 | 9
  Any HIV (Month 12.5) | 0.172 [0.127 to 0.209] | 0.314 [0.165 to 0.526] | 0.148 [0.112 to 0.263] | 0.188 [0.125 to 0.252]
  Env ZM96 (Month 12.5): number analyzed (Participants) | 15 | 20 | 6 | 8
  Env ZM96 (Month 12.5) | 0.149 [0.077 to 0.248] | 0.172 [0.124 to 0.288] | 0.202 [0.146 to 0.242] | 0.126 [0.099 to 0.201]
  Env-1-ZM96 (Month 12.5): number analyzed (Participants) | 15 | 20 | 5 | 9
  Env-1-ZM96 (Month 12.5) | 0.14 [0.092 to 0.257] | 0.135 [0.099 to 0.183] | 0.157 [0.098 to 0.173] | 0.106 [0.096 to 0.206]
  Env-2-ZM96 (Month 12.5): number analyzed (Participants) | 1 | 8 | 4 | 0
  Env-2-ZM96 (Month 12.5) | 0.128 [0.128 to 0.128] | 0.163 [0.087 to 0.258] | 0.084 [0.075 to 0.094] |
  LAI Gag (Month 12.5): number analyzed (Participants) | 1 | 2 | 1 | 1
  LAI Gag (Month 12.5) | 0.11 [0.11 to 0.11] | 0.085 [0.071 to 0.099] | 0.136 [0.136 to 0.136] | 0.081 [0.081 to 0.081]
  TV1 gp120 (Month 12.5): number analyzed (Participants) | 20 | 24 | 16 | 8
  TV1 gp120 (Month 12.5) | 0.133 [0.103 to 0.228] | 0.275 [0.138 to 0.379] | 0.138 [0.112 to 0.233] | 0.147 [0.1 to 0.236]
  1086 gp120 (Month 18): number analyzed (Participants) | 9 | 21 | 10 | 5
  1086 gp120 (Month 18) | 0.106 [0.095 to 0.126] | 0.121 [0.093 to 0.237] | 0.121 [0.099 to 0.133] | 0.107 [0.089 to 0.116]
  Any Env (Month 18): number analyzed (Participants) | 16 | 23 | 13 | 9
  Any Env (Month 18) | 0.117 [0.082 to 0.19] | 0.169 [0.096 to 0.272] | 0.122 [0.121 to 0.157] | 0.123 [0.085 to 0.164]
  Any HIV (Month 18): number analyzed (Participants) | 17 | 23 | 14 | 9
  Any HIV (Month 18) | 0.105 [0.079 to 0.186] | 0.156 [0.115 to 0.329] | 0.129 [0.102 to 0.178] | 0.123 [0.115 to 0.187]
  Env ZM96 (Month 18): number analyzed (Participants) | 14 | 18 | 4 | 6
  Env ZM96 (Month 18) | 0.085 [0.062 to 0.132] | 0.133 [0.087 to 0.155] | 0.117 [0.114 to 0.121] | 0.133 [0.093 to 0.165]
  Env-1-ZM96 (Month 18): number analyzed (Participants) | 14 | 20 | 3 | 6
  Env-1-ZM96 (Month 18) | 0.09 [0.07 to 0.131] | 0.111 [0.078 to 0.131] | 0.077 [0.072 to 0.083] | 0.124 [0.081 to 0.14]
  Env-2-ZM96 (Month 18): number analyzed (Participants) | 0 | 4 | 2 | 0
  Env-2-ZM96 (Month 18) |  | 0.132 [0.118 to 0.175] | 0.064 [0.055 to 0.072] |
  LAI Gag (Month 18): number analyzed (Participants) | 1 | 2 | 1 | 0
  LAI Gag (Month 18) | 0.076 [0.076 to 0.076] | 0.059 [0.051 to 0.067] | 0.07 [0.07 to 0.07] |
  TV1 gp120 (Month 18): number analyzed (Participants) | 11 | 23 | 11 | 7
  TV1 gp120 (Month 18) | 0.109 [0.084 to 0.217] | 0.158 [0.105 to 0.258] | 0.122 [0.11 to 0.168] | 0.085 [0.076 to 0.113]

27. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG3 Ab Binding to Env Proteins
Description: Serum IgG3 responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:40 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if they meet three criteria: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI.
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 31 | 29 | 33 | 18
Participants
  1086C_D7gp120.avi/293F (Month 6.5): number analyzed (Participants) | 30 | 28 | 33 | 18
  1086C_D7gp120.avi/293F (Month 6.5) | 28 | 27 | 30 | 18
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 31 | 28 | 33 | 18
  96ZM651.D11gp120.avi (Month 6.5) | 27 | 24 | 26 | 16
  AE.A244 V1V2 Tags/293F (Month 6.5): number analyzed (Participants) | 30 | 26 | 33 | 17
  AE.A244 V1V2 Tags/293F (Month 6.5) | 9 | 13 | 14 | 3
  C.1086C_V1_V2 Tags (Month 6.5): number analyzed (Participants) | 30 | 27 | 32 | 17
  C.1086C_V1_V2 Tags (Month 6.5) | 9 | 12 | 13 | 2
  Con 6 gp120/B (Month 6.5): number analyzed (Participants) | 30 | 28 | 33 | 18
  Con 6 gp120/B (Month 6.5) | 19 | 22 | 18 | 15
  Con S gp140 CFI (Month 6.5): number analyzed (Participants) | 30 | 28 | 33 | 18
  Con S gp140 CFI (Month 6.5) | 28 | 27 | 25 | 17
  TV1c8_D11gp120.avi/293F (Month 6.5): number analyzed (Participants) | 30 | 27 | 33 | 18
  TV1c8_D11gp120.avi/293F (Month 6.5) | 27 | 26 | 29 | 17
  gp41 (Month 6.5): number analyzed (Participants) | 31 | 28 | 32 | 17
  gp41 (Month 6.5) | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 6.5): number analyzed (Participants) | 29 | 27 | 31 | 16
  gp70-96ZM651.02 V1v2 (Month 6.5) | 2 | 3 | 7 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 30 | 28 | 32 | 16
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 3 | 3 | 10 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 30 | 28 | 32 | 16
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 3 | 3 | 7 | 0
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 30 | 28 | 32 | 16
  gp70_B.CaseA_V1_V2 (Month 6.5) | 2 | 2 | 7 | 0
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 31 | 28 | 31 | 17
  1086C_D7gp120.avi/293F (Month 12) | 11 | 16 | 17 | 8
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 31 | 28 | 31 | 17
  96ZM651.D11gp120.avi (Month 12) | 0 | 2 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 30 | 28 | 31 | 16
  AE.A244 V1V2 Tags/293F (Month 12) | 1 | 0 | 2 | 0
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 30 | 28 | 31 | 16
  C.1086C_V1_V2 Tags (Month 12) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 31 | 28 | 31 | 17
  Con 6 gp120/B (Month 12) | 0 | 0 | 0 | 0
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 31 | 28 | 31 | 17
  Con S gp140 CFI (Month 12) | 1 | 2 | 1 | 0
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 31 | 28 | 31 | 17
  TV1c8_D11gp120.avi/293F (Month 12) | 3 | 3 | 5 | 2
  gp41 (Month 12): number analyzed (Participants) | 31 | 28 | 29 | 16
  gp41 (Month 12) | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 12): number analyzed (Participants) | 29 | 28 | 29 | 15
  gp70-96ZM651.02 V1v2 (Month 12) | 1 | 0 | 1 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 30 | 28 | 30 | 15
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 1 | 0 | 1 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 30 | 28 | 30 | 15
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 1 | 1 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 30 | 28 | 30 | 15
  gp70_B.CaseA_V1_V2 (Month 12) | 1 | 0 | 0 | 0
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  1086C_D7gp120.avi/293F (Month 12.5) | 28 | 28 | 29 | 15
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  96ZM651.D11gp120.avi (Month 12.5) | 14 | 17 | 14 | 8
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 16
  AE.A244 V1V2 Tags/293F (Month 12.5) | 6 | 9 | 13 | 4
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 16
  C.1086C_V1_V2 Tags (Month 12.5) | 4 | 7 | 10 | 1
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  Con 6 gp120/B (Month 12.5) | 6 | 10 | 5 | 4
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  Con S gp140 CFI (Month 12.5) | 18 | 21 | 19 | 10
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  TV1c8_D11gp120.avi/293F (Month 12.5) | 25 | 25 | 28 | 13
  gp41 (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 16
  gp41 (Month 12.5) | 0 | 0 | 0 | 1
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 30 | 29 | 29 | 15
  gp70-96ZM651.02 V1v2 (Month 12.5) | 3 | 3 | 5 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 2 | 2 | 8 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 1 | 2 | 7 | 0
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70_B.CaseA_V1_V2 (Month 12.5) | 1 | 2 | 4 | 0
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  1086C_D7gp120.avi/293F (Month 18) | 11 | 16 | 15 | 4
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  96ZM651.D11gp120.avi (Month 18) | 0 | 0 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 15
  AE.A244 V1V2 Tags/293F (Month 18) | 1 | 0 | 5 | 0
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 15
  C.1086C_V1_V2 Tags (Month 18) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  Con 6 gp120/B (Month 18) | 0 | 0 | 1 | 0
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  Con S gp140 CFI (Month 18) | 4 | 4 | 0 | 0
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  TV1c8_D11gp120.avi/293F (Month 18) | 6 | 6 | 4 | 2
  gp41 (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 15
  gp41 (Month 18) | 0 | 0 | 0 | 2
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 28 | 29 | 30 | 14
  gp70-96ZM651.02 V1v2 (Month 18) | 1 | 0 | 2 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 1 | 0 | 1 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 1 | 0 | 1 | 0
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70_B.CaseA_V1_V2 (Month 18) | 1 | 0 | 0 | 0

28. Secondary Outcome: Level of Vaccine-induced Serum IgG3 Ab Binding to Env Proteins
Description: Serum IgG3 responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:40 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Summary was calculated among positive responders only (positivity criteria are described in Outcome 1).
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 28 | 28 | 30 | 18
relative fluorescence units
  1086C_D7gp120.avi/293F (Month 6.5): number analyzed (Participants) | 28 | 27 | 30 | 18
  1086C_D7gp120.avi/293F (Month 6.5) | 3002.2 [1394.2 to 5955.3] | 3236 [2115.9 to 8234.4] | 2824 [1284.9 to 4232.1] | 2728.9 [1994.4 to 5368.3]
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 27 | 24 | 26 | 16
  96ZM651.D11gp120.avi (Month 6.5) | 810.5 [364.6 to 2145.9] | 594.5 [318.3 to 1383.3] | 448.1 [315.6 to 1256.3] | 613.2 [299.9 to 965.6]
  AE.A244 V1V2 Tags/293F (Month 6.5): number analyzed (Participants) | 9 | 13 | 14 | 3
  AE.A244 V1V2 Tags/293F (Month 6.5) | 596.8 [267.8 to 1343.5] | 265 [162.2 to 547.5] | 527.2 [338.8 to 1143.7] | 135.2 [128.5 to 350.6]
  C.1086C_V1_V2 Tags (Month 6.5): number analyzed (Participants) | 9 | 12 | 13 | 2
  C.1086C_V1_V2 Tags (Month 6.5) | 372.2 [154.5 to 885] | 218.4 [135.9 to 409.5] | 418.8 [274.8 to 1135.8] | 222.1 [173.3 to 270.9]
  Con 6 gp120/B (Month 6.5): number analyzed (Participants) | 19 | 22 | 18 | 15
  Con 6 gp120/B (Month 6.5) | 384.2 [256.2 to 619.1] | 299.2 [222.2 to 645.2] | 260.6 [168.3 to 431.9] | 197.2 [147.8 to 232.1]
  Con S gp140 CFI (Month 6.5): number analyzed (Participants) | 28 | 27 | 25 | 17
  Con S gp140 CFI (Month 6.5) | 653.1 [413.8 to 1959.5] | 936.8 [534.8 to 2301.9] | 497.8 [320 to 1017] | 435.2 [346.5 to 885]
  TV1c8_D11gp120.avi/293F (Month 6.5): number analyzed (Participants) | 27 | 26 | 29 | 17
  TV1c8_D11gp120.avi/293F (Month 6.5) | 2134.8 [494 to 4958.9] | 1517.2 [618.8 to 2555.9] | 1306.2 [665 to 3785.2] | 2277 [1024.2 to 3621]
  gp41 (Month 6.5): number analyzed (Participants) | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 6.5): number analyzed (Participants) | 2 | 3 | 7 | 0
  gp70-96ZM651.02 V1v2 (Month 6.5) | 3929.5 [2035.8 to 5823.2] | 790 [536 to 898.8] | 1142 [760.2 to 1352.5] |
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 3 | 3 | 10 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 3242.8 [1691.4 to 5474.6] | 230.2 [223.8 to 407.2] | 512.6 [177.4 to 1562.3] |
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 3 | 3 | 7 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 501.8 [339 to 6053.9] | 257.5 [250.9 to 440.6] | 1197 [473.6 to 1605] |
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 2 | 2 | 7 | 0
  gp70_B.CaseA_V1_V2 (Month 6.5) | 4118.6 [2113.9 to 6123.3] | 742 [498.8 to 985.2] | 858.5 [134.6 to 2379.6] |
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 11 | 16 | 17 | 8
  1086C_D7gp120.avi/293F (Month 12) | 327 [195.5 to 453.1] | 288.8 [203.6 to 805.1] | 164.5 [121.8 to 301.2] | 220.4 [150.2 to 365.7]
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 0 | 2 | 0 | 0
  96ZM651.D11gp120.avi (Month 12) |  | 131.5 [129.2 to 133.8] |  |
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 1 | 0 | 2 | 0
  AE.A244 V1V2 Tags/293F (Month 12) | 148.2 [148.2 to 148.2] |  | 605.9 [363.3 to 848.4] |
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 0
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 1 | 2 | 1 | 0
  Con S gp140 CFI (Month 12) | 297.8 [297.8 to 297.8] | 100.4 [100.2 to 100.6] | 125.8 [125.8 to 125.8] |
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 3 | 3 | 5 | 2
  TV1c8_D11gp120.avi/293F (Month 12) | 128.8 [118.9 to 2735.2] | 148.8 [129.4 to 168] | 281.5 [236 to 1467.5] | 9282.5 [5013.1 to 13551.9]
  gp41 (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 12): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70-96ZM651.02 V1v2 (Month 12) | 502.8 [502.8 to 502.8] |  | 268.8 [268.8 to 268.8] |
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 874.8 [874.8 to 874.8] |  | 121.8 [121.8 to 121.8] |
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 1 | 1 | 0 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 1348.5 [1348.5 to 1348.5] | 225 [225 to 225] |  |
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 12) | 798.2 [798.2 to 798.2] |  |  |
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 28 | 28 | 29 | 15
  1086C_D7gp120.avi/293F (Month 12.5) | 1049.2 [390 to 2565.1] | 1184.2 [711.1 to 3716.6] | 1086.2 [606.8 to 2699.8] | 1739 [593.4 to 5582.2]
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 14 | 17 | 14 | 8
  96ZM651.D11gp120.avi (Month 12.5) | 300.9 [161.9 to 838.8] | 314.5 [149 to 681.5] | 314.9 [189.6 to 439.3] | 264.5 [203.9 to 391]
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 6 | 9 | 13 | 4
  AE.A244 V1V2 Tags/293F (Month 12.5) | 283.9 [178.3 to 762] | 271 [193.5 to 666.2] | 480 [289.2 to 697] | 479.1 [308.5 to 5950.9]
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 4 | 7 | 10 | 1
  C.1086C_V1_V2 Tags (Month 12.5) | 470 [320.7 to 1060.8] | 197.8 [152.6 to 332.5] | 379.2 [218.2 to 473] | 22000 [22000 to 22000]
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 6 | 10 | 5 | 4
  Con 6 gp120/B (Month 12.5) | 284 [197.3 to 345.2] | 329.5 [174.1 to 376] | 540 [278.5 to 672.5] | 203 [131 to 510.4]
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 18 | 21 | 19 | 10
  Con S gp140 CFI (Month 12.5) | 264.1 [179 to 623.1] | 322.8 [202.2 to 1225.2] | 208.2 [160.5 to 382.6] | 476.8 [118.7 to 581.4]
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 25 | 25 | 28 | 13
  TV1c8_D11gp120.avi/293F (Month 12.5) | 586.8 [385.5 to 2959.5] | 673.8 [415 to 2072.2] | 439.4 [199.9 to 1111.1] | 1017.2 [708 to 3056.2]
  gp41 (Month 12.5): number analyzed (Participants) | 0 | 0 | 0 | 1
  gp41 (Month 12.5) |  |  |  | 3020.8 [3020.8 to 3020.8]
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 3 | 3 | 5 | 1
  gp70-96ZM651.02 V1v2 (Month 12.5) | 157.8 [130.9 to 992.2] | 354 [287.8 to 431.9] | 2402.8 [1323.5 to 3308.5] | 4707.5 [4707.5 to 4707.5]
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 2 | 2 | 8 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 853.5 [564.1 to 1142.9] | 231.6 [181.9 to 281.3] | 487.8 [167.2 to 1114.6] |
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 1 | 2 | 7 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 2010.8 [2010.8 to 2010.8] | 255.4 [191.4 to 319.3] | 551 [175 to 850.4] |
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 1 | 2 | 4 | 0
  gp70_B.CaseA_V1_V2 (Month 12.5) | 1262.5 [1262.5 to 1262.5] | 233.5 [205.1 to 261.9] | 1457.8 [642 to 2307.9] |
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 11 | 16 | 15 | 4
  1086C_D7gp120.avi/293F (Month 18) | 204 [146.2 to 522.4] | 266.4 [172.9 to 555.9] | 167.5 [158.5 to 217.5] | 133 [109.4 to 236.1]
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 1 | 0 | 5 | 0
  AE.A244 V1V2 Tags/293F (Month 18) | 187.8 [187.8 to 187.8] |  | 245.2 [197.2 to 479.5] |
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 0 | 0 | 1 | 0
  Con 6 gp120/B (Month 18) |  |  | 368.8 [368.8 to 368.8] |
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 4 | 4 | 0 | 0
  Con S gp140 CFI (Month 18) | 126.6 [100 to 155.2] | 136.6 [126.4 to 156.8] |  |
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 6 | 6 | 4 | 2
  TV1c8_D11gp120.avi/293F (Month 18) | 451.2 [202.6 to 915.9] | 198.9 [125.4 to 362] | 725.9 [239.6 to 1298.6] | 6535.8 [3329.8 to 9741.8]
  gp41 (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 2
  gp41 (Month 18) |  |  |  | 9170.6 [6114.3 to 12226.9]
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 1 | 0 | 2 | 0
  gp70-96ZM651.02 V1v2 (Month 18) | 434.8 [434.8 to 434.8] |  | 196.6 [151.1 to 242.2] |
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 534.8 [534.8 to 534.8] |  | 170.5 [170.5 to 170.5] |
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 887.5 [887.5 to 887.5] |  | 177.5 [177.5 to 177.5] |
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 18) | 474 [474 to 474] |  |  |

29. Secondary Outcome: Occurrence of Vaccine-induced Serum IgA Ab Binding to Env Proteins
Description: as for outcome 3
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 28 | 25 | 30 | 17
Participants
  00MSA 4076 gp140 (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 17
  00MSA 4076 gp140 (Month 6.5) | 10 | 11 | 17 | 5
  1086C_D7gp120.avi/293F (Month 6.5): number analyzed (Participants) | 24 | 20 | 29 | 16
  1086C_D7gp120.avi/293F (Month 6.5) | 22 | 19 | 27 | 14
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 16
  96ZM651.D11gp120.avi (Month 6.5) | 12 | 8 | 22 | 4
  A1.con.env03 140 CF (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 17
  A1.con.env03 140 CF (Month 6.5) | 11 | 8 | 18 | 6
  AE.A244 V1V2 Tags/293F (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 17
  AE.A244 V1V2 Tags/293F (Month 6.5) | 1 | 0 | 1 | 1
  C.1086C_V1_V2 Tags (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 17
  C.1086C_V1_V2 Tags (Month 6.5) | 1 | 1 | 1 | 1
  Con 6 gp120/B (Month 6.5): number analyzed (Participants) | 25 | 24 | 30 | 17
  Con 6 gp120/B (Month 6.5) | 10 | 9 | 15 | 4
  Con S gp140 CFI (Month 6.5): number analyzed (Participants) | 25 | 24 | 30 | 17
  Con S gp140 CFI (Month 6.5) | 17 | 16 | 24 | 7
  TV1c8_D11gp120.avi/293F (Month 6.5): number analyzed (Participants) | 25 | 24 | 29 | 17
  TV1c8_D11gp120.avi/293F (Month 6.5) | 18 | 19 | 27 | 11
  gp41 (Month 6.5): number analyzed (Participants) | 26 | 24 | 30 | 17
  gp41 (Month 6.5) | 0 | 1 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 6.5): number analyzed (Participants) | 24 | 22 | 26 | 15
  gp70-96ZM651.02 V1v2 (Month 6.5) | 0 | 0 | 0 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 24 | 22 | 26 | 14
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 1 | 0 | 0 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 24 | 22 | 26 | 15
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 1 | 0 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 24 | 21 | 26 | 15
  gp70_B.CaseA_V1_V2 (Month 6.5) | 0 | 0 | 0 | 0
  00MSA 4076 gp140 (Month 12): number analyzed (Participants) | 28 | 25 | 28 | 17
  00MSA 4076 gp140 (Month 12) | 3 | 3 | 4 | 1
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 26 | 21 | 27 | 16
  1086C_D7gp120.avi/293F (Month 12) | 20 | 17 | 24 | 11
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 28 | 25 | 28 | 16
  96ZM651.D11gp120.avi (Month 12) | 2 | 4 | 4 | 1
  A1.con.env03 140 CF (Month 12): number analyzed (Participants) | 28 | 25 | 28 | 17
  A1.con.env03 140 CF (Month 12) | 3 | 3 | 5 | 1
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 28 | 25 | 28 | 17
  AE.A244 V1V2 Tags/293F (Month 12) | 1 | 0 | 0 | 0
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 27 | 25 | 28 | 17
  C.1086C_V1_V2 Tags (Month 12) | 1 | 0 | 0 | 0
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 26 | 25 | 28 | 16
  Con 6 gp120/B (Month 12) | 3 | 2 | 3 | 1
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 27 | 25 | 28 | 17
  Con S gp140 CFI (Month 12) | 4 | 4 | 7 | 2
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 27 | 25 | 27 | 17
  TV1c8_D11gp120.avi/293F (Month 12) | 7 | 10 | 22 | 5
  gp41 (Month 12): number analyzed (Participants) | 28 | 25 | 28 | 17
  gp41 (Month 12) | 0 | 0 | 0 | 0
  gp70-96ZM651.02 V1v2 (Month 12): number analyzed (Participants) | 25 | 22 | 23 | 16
  gp70-96ZM651.02 V1v2 (Month 12) | 0 | 0 | 0 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 25 | 23 | 23 | 15
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 1 | 1 | 0 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 25 | 23 | 23 | 16
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 1 | 0 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 25 | 23 | 23 | 16
  gp70_B.CaseA_V1_V2 (Month 12) | 0 | 1 | 0 | 0

30. Secondary Outcome: Level of Vaccine-induced Serum IgA Ab Binding to Env Proteins
Description: Serum IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:10 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI < 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Summary was calculated among positive responders only (positivity criteria are described in Outcome 1).
Time Frame: Measured at Months 6.5 and 12.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 22 | 19 | 27 | 14
relative fluorescence units
  00MSA 4076 gp140 (Month 6.5): number analyzed (Participants) | 10 | 11 | 17 | 5
  00MSA 4076 gp140 (Month 6.5) | 1845.2 [488.2 to 8688.9] | 661 [255.5 to 1376.9] | 1434.2 [526.8 to 8249.5] | 2502 [1231.5 to 2833.8]
  1086C_D7gp120.avi/293F (Month 6.5) | 22000 [17472 to 22000] | 22000 [13255.1 to 22000] | 22000 [22000 to 22000] | 20863 [11859 to 22000]
  96ZM651.D11gp120.avi (Month 6.5): number analyzed (Participants) | 12 | 8 | 22 | 4
  96ZM651.D11gp120.avi (Month 6.5) | 8047.1 [6816.6 to 13252.6] | 8849.6 [6323.8 to 10004.8] | 7595.5 [5318.3 to 13822.1] | 11444 [7878.1 to 15391.1]
  A1.con.env03 140 CF (Month 6.5): number analyzed (Participants) | 11 | 8 | 18 | 6
  A1.con.env03 140 CF (Month 6.5) | 2823.8 [535.9 to 8015.5] | 1407.1 [612.2 to 1760.2] | 1909.9 [648.1 to 6867.4] | 2191.9 [1343.3 to 5852.8]
  AE.A244 V1V2 Tags/293F (Month 6.5): number analyzed (Participants) | 1 | 0 | 1 | 1
  AE.A244 V1V2 Tags/293F (Month 6.5) | 6260.8 [6260.8 to 6260.8] |  | 1998 [1998 to 1998] | 4791.2 [4791.2 to 4791.2]
  C.1086C_V1_V2 Tags (Month 6.5): number analyzed (Participants) | 1 | 1 | 1 | 1
  C.1086C_V1_V2 Tags (Month 6.5) | 9201.2 [9201.2 to 9201.2] | 882.5 [882.5 to 882.5] | 1978.5 [1978.5 to 1978.5] | 4818.8 [4818.8 to 4818.8]
  Con 6 gp120/B (Month 6.5): number analyzed (Participants) | 10 | 9 | 15 | 4
  Con 6 gp120/B (Month 6.5) | 9493.6 [3152.8 to 11729.6] | 3719.8 [3271.2 to 4214] | 4863.5 [3355.6 to 7182] | 6432.1 [3135 to 9692.9]
  Con S gp140 CFI (Month 6.5): number analyzed (Participants) | 17 | 16 | 24 | 7
  Con S gp140 CFI (Month 6.5) | 5888.5 [3208.2 to 17024.2] | 4698.9 [3204.9 to 6151.9] | 6925.8 [3836.3 to 22000] | 5943.2 [4851.8 to 13324]
  TV1c8_D11gp120.avi/293F (Month 6.5): number analyzed (Participants) | 18 | 19 | 27 | 11
  TV1c8_D11gp120.avi/293F (Month 6.5) | 8312.8 [3759.4 to 19844.6] | 5613.2 [1829.4 to 7662.5] | 12210.8 [6345.9 to 22000] | 4144.5 [3052.5 to 13847.4]
  gp41 (Month 6.5): number analyzed (Participants) | 0 | 1 | 0 | 0
  gp41 (Month 6.5) |  | 3047.2 [3047.2 to 3047.2] |  |
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 813.8 [813.8 to 813.8] |  |  |
  gp70_B.CaseA2 V1/V2/169K (Month 6.5): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 6.5) | 22000 [22000 to 22000] |  |  |
  gp70_B.CaseA_V1_V2 (Month 6.5): number analyzed (Participants) | 0 | 0 | 0 | 0
  00MSA 4076 gp140 (Month 12): number analyzed (Participants) | 3 | 3 | 4 | 1
  00MSA 4076 gp140 (Month 12) | 2229 [1760 to 5844.8] | 1486.5 [813.4 to 2417] | 1501.5 [421.4 to 3012.2] | 727.5 [727.5 to 727.5]
  1086C_D7gp120.avi/293F (Month 12): number analyzed (Participants) | 20 | 17 | 24 | 11
  1086C_D7gp120.avi/293F (Month 12) | 7533.6 [4651.4 to 16946] | 4962.8 [2254.8 to 7956.5] | 9267.8 [5751.8 to 15500.5] | 3780.8 [2303.6 to 9670.9]
  96ZM651.D11gp120.avi (Month 12): number analyzed (Participants) | 2 | 4 | 4 | 1
  96ZM651.D11gp120.avi (Month 12) | 5390.6 [4675.2 to 6106.1] | 10692 [8753.4 to 13069.9] | 6160 [5252.9 to 7161.4] | 10678.8 [10678.8 to 10678.8]
  A1.con.env03 140 CF (Month 12): number analyzed (Participants) | 3 | 3 | 5 | 1
  A1.con.env03 140 CF (Month 12) | 6053.5 [3152.1 to 6928.8] | 2047.2 [1493.4 to 2679.6] | 1051.8 [580.2 to 7617] | 1290 [1290 to 1290]
  AE.A244 V1V2 Tags/293F (Month 12): number analyzed (Participants) | 1 | 0 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 12) | 3551 [3551 to 3551] |  |  |
  C.1086C_V1_V2 Tags (Month 12): number analyzed (Participants) | 1 | 0 | 0 | 0
  C.1086C_V1_V2 Tags (Month 12) | 6647 [6647 to 6647] |  |  |
  Con 6 gp120/B (Month 12): number analyzed (Participants) | 3 | 2 | 3 | 1
  Con 6 gp120/B (Month 12) | 3134.5 [2691.1 to 3441.2] | 5267.4 [4380.6 to 6154.2] | 2058 [2014 to 3017.9] | 3144 [3144 to 3144]
  Con S gp140 CFI (Month 12): number analyzed (Participants) | 4 | 4 | 7 | 2
  Con S gp140 CFI (Month 12) | 5268 [2966.7 to 10882.8] | 7882.6 [2290.9 to 15009.9] | 5614.8 [3224.8 to 12063.2] | 5104.8 [4650.4 to 5559.1]
  TV1c8_D11gp120.avi/293F (Month 12): number analyzed (Participants) | 7 | 10 | 22 | 5
  TV1c8_D11gp120.avi/293F (Month 12) | 3505.5 [1538.2 to 4408.2] | 1366.6 [875.6 to 2180.6] | 2812 [1200.9 to 6530.2] | 4003 [2953.5 to 14074.2]
  gp41 (Month 12): number analyzed (Participants) | 0 | 0 | 0 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12): number analyzed (Participants) | 1 | 1 | 0 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12) | 137.5 [137.5 to 137.5] | 993 [993 to 993] |  |
  gp70_B.CaseA2 V1/V2/169K (Month 12): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12) | 22000 [22000 to 22000] |  |  |
  gp70_B.CaseA_V1_V2 (Month 12): number analyzed (Participants) | 0 | 1 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 12) |  | 1540 [1540 to 1540] |  |

31. Secondary Outcome: HIV-specific CD4+ T Cell Polyfunctionality by ICS - Functionality Scores
Description: COMPASS uses a Bayesian hierarchical framework to model all observed functional cell subsets and select those most likely to exhibit antigen-specific responses. Cell-subset responses are quantified by posterior probabilities. The functionality score (FS) summarizes, as a single number for each participant, the proportion of antigen-specific cell subsets among all measured subsets, irrespective of degree of functionality. FS ranges from zero to one. FS will assign a higher score to participants that exhibit antigen specificity in more cell subsets irrespective of their degree of functionality.
Time Frame: Measured at Months 6.5, 12, 12.5, and 18
Population: "Overall Number of Participants Analyzed" represents the number of participants in the per-protocol population. "Number Analyzed" shows the number of HIV uninfected participants with available COMPASS data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: Functionality Score
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 27 | 30 | 31 | 19
Functionality Score
  1086 gp120 (Month 6.5): number analyzed (Participants) | 25 | 26 | 26 | 15
  1086 gp120 (Month 6.5) | 0.169 [0.108 to 0.204] | 0.171 [0.147 to 0.217] | 0.158 [0.136 to 0.2] | 0.15 [0.13 to 0.18]
  1086 gp120 (Month 12): number analyzed (Participants) | 26 | 29 | 27 | 17
  1086 gp120 (Month 12) | 0.108 [0.069 to 0.148] | 0.129 [0.111 to 0.161] | 0.129 [0.084 to 0.16] | 0.101 [0.076 to 0.12]
  1086 gp120 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  1086 gp120 (Month 12.5) | 0.17 [0.148 to 0.206] | 0.188 [0.149 to 0.229] | 0.131 [0.087 to 0.173] | 0.138 [0.097 to 0.191]
  1086 gp120 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  1086 gp120 (Month 18) | 0.143 [0.118 to 0.185] | 0.156 [0.126 to 0.179] | 0.111 [0.079 to 0.165] | 0.114 [0.091 to 0.139]
  Any Env ZM96 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  Any Env ZM96 (Month 6.5) | 0.157 [0.109 to 0.21] | 0.175 [0.116 to 0.203] | 0.126 [0.094 to 0.155] | 0.123 [0.078 to 0.193]
  Any Env ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Any Env ZM96 (Month 12) | 0.126 [0.085 to 0.166] | 0.129 [0.115 to 0.159] | 0.106 [0.068 to 0.13] | 0.111 [0.093 to 0.15]
  Any Env ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Any Env ZM96 (Month 12.5) | 0.187 [0.12 to 0.225] | 0.197 [0.142 to 0.224] | 0.117 [0.087 to 0.144] | 0.158 [0.12 to 0.183]
  Any Env ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Any Env ZM96 (Month 18) | 0.159 [0.089 to 0.179] | 0.163 [0.112 to 0.181] | 0.11 [0.083 to 0.128] | 0.131 [0.054 to 0.157]
  Env-1-ZM96 (Month 6.5): number analyzed (Participants) | 27 | 26 | 28 | 17
  Env-1-ZM96 (Month 6.5) | 0.157 [0.109 to 0.21] | 0.177 [0.119 to 0.203] | 0.126 [0.094 to 0.155] | 0.123 [0.078 to 0.193]
  Env-1-ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Env-1-ZM96 (Month 12) | 0.126 [0.085 to 0.166] | 0.129 [0.115 to 0.159] | 0.106 [0.068 to 0.124] | 0.111 [0.093 to 0.15]
  Env-1-ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Env-1-ZM96 (Month 12.5) | 0.187 [0.12 to 0.225] | 0.197 [0.142 to 0.224] | 0.117 [0.087 to 0.144] | 0.158 [0.12 to 0.183]
  Env-1-ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Env-1-ZM96 (Month 18) | 0.159 [0.089 to 0.179] | 0.163 [0.112 to 0.181] | 0.11 [0.082 to 0.128] | 0.131 [0.054 to 0.157]
  Env-2-ZM96 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  Env-2-ZM96 (Month 6.5) | 0.032 [0.015 to 0.072] | 0.027 [0.017 to 0.076] | 0.04 [0.028 to 0.068] | 0.046 [0.023 to 0.062]
  Env-2-ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Env-2-ZM96 (Month 12) | 0.015 [0.003 to 0.024] | 0.044 [0.015 to 0.074] | 0.032 [0.011 to 0.072] | 0.033 [0.018 to 0.047]
  Env-2-ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Env-2-ZM96 (Month 12.5) | 0.024 [0.013 to 0.061] | 0.065 [0.022 to 0.098] | 0.023 [0.018 to 0.038] | 0.033 [0.013 to 0.071]
  Env-2-ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Env-2-ZM96 (Month 18) | 0.016 [0.007 to 0.026] | 0.039 [0.019 to 0.082] | 0.021 [0.011 to 0.062] | 0.028 [0.011 to 0.039]
  LAI-Gag (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  LAI-Gag (Month 6.5) | 0.04 [0.021 to 0.069] | 0.057 [0.027 to 0.071] | 0.03 [0.012 to 0.039] | 0.036 [0.029 to 0.069]
  LAI-Gag (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  LAI-Gag (Month 12) | 0.04 [0.014 to 0.053] | 0.04 [0.015 to 0.066] | 0.025 [0.009 to 0.042] | 0.026 [0.016 to 0.05]
  LAI-Gag (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  LAI-Gag (Month 12.5) | 0.03 [0.016 to 0.07] | 0.041 [0.02 to 0.069] | 0.037 [0.023 to 0.055] | 0.038 [0.012 to 0.068]
  LAI-Gag (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  LAI-Gag (Month 18) | 0.024 [0.016 to 0.041] | 0.031 [0.018 to 0.065] | 0.02 [0.011 to 0.038] | 0.037 [0.017 to 0.061]
  TV1 gp120 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  TV1 gp120 (Month 6.5) | 0.165 [0.122 to 0.227] | 0.186 [0.143 to 0.214] | 0.177 [0.137 to 0.218] | 0.156 [0.121 to 0.187]
  TV1 gp120 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  TV1 gp120 (Month 12) | 0.125 [0.105 to 0.179] | 0.165 [0.107 to 0.192] | 0.153 [0.112 to 0.178] | 0.124 [0.065 to 0.145]
  TV1 gp120 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  TV1 gp120 (Month 12.5) | 0.217 [0.173 to 0.232] | 0.231 [0.161 to 0.252] | 0.172 [0.125 to 0.207] | 0.15 [0.113 to 0.205]
  TV1 gp120 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  TV1 gp120 (Month 18) | 0.161 [0.136 to 0.21] | 0.172 [0.16 to 0.199] | 0.143 [0.119 to 0.177] | 0.099 [0.055 to 0.17]

32. Secondary Outcome: HIV-specific CD4+ T Cell Polyfunctionality by ICS - Polyfunctionality Scores
Description: COMPASS uses a Bayesian hierarchical framework to model all observed functional cell subsets and select those most likely to exhibit antigen-specific responses. Cell-subset responses are quantified by posterior probabilities. The polyfunctionality score (PFS) summarizes, as a single number for each participant, the proportion of antigen-specific cell subsets among all measured subsets, weighted by the degree of functionality of the corresponding subset. PFS ranges from zero to one. PFS will assign a higher score to participants with antigen-specific cell subsets of higher degree.
Time Frame: Measured at Months 6.5, 12, 12.5, and 18
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: Polyfunctionality Score
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 27 | 30 | 31 | 19
Polyfunctionality Score
  1086 gp120 (Month 6.5): number analyzed (Participants) | 25 | 26 | 26 | 15
  1086 gp120 (Month 6.5) | 0.11 [0.051 to 0.135] | 0.12 [0.095 to 0.141] | 0.098 [0.065 to 0.122] | 0.106 [0.09 to 0.116]
  1086 gp120 (Month 12): number analyzed (Participants) | 26 | 29 | 27 | 17
  1086 gp120 (Month 12) | 0.067 [0.05 to 0.105] | 0.087 [0.064 to 0.113] | 0.062 [0.049 to 0.098] | 0.07 [0.038 to 0.081]
  1086 gp120 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  1086 gp120 (Month 12.5) | 0.108 [0.076 to 0.135] | 0.129 [0.082 to 0.148] | 0.067 [0.048 to 0.098] | 0.091 [0.053 to 0.109]
  1086 gp120 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  1086 gp120 (Month 18) | 0.1 [0.072 to 0.121] | 0.108 [0.08 to 0.126] | 0.062 [0.044 to 0.099] | 0.064 [0.056 to 0.09]
  Any Env ZM96 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  Any Env ZM96 (Month 6.5) | 0.111 [0.084 to 0.134] | 0.124 [0.091 to 0.136] | 0.083 [0.051 to 0.105] | 0.092 [0.058 to 0.124]
  Any Env ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Any Env ZM96 (Month 12) | 0.082 [0.063 to 0.119] | 0.099 [0.062 to 0.107] | 0.06 [0.042 to 0.086] | 0.09 [0.049 to 0.101]
  Any Env ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Any Env ZM96 (Month 12.5) | 0.127 [0.087 to 0.146] | 0.132 [0.088 to 0.144] | 0.069 [0.046 to 0.09] | 0.111 [0.088 to 0.12]
  Any Env ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Any Env ZM96 (Month 18) | 0.114 [0.064 to 0.127] | 0.115 [0.083 to 0.126] | 0.066 [0.042 to 0.095] | 0.085 [0.046 to 0.111]
  Env-1-ZM96 (Month 6.5): number analyzed (Participants) | 27 | 26 | 28 | 17
  Env-1-ZM96 (Month 6.5) | 0.111 [0.084 to 0.134] | 0.124 [0.094 to 0.136] | 0.083 [0.051 to 0.105] | 0.092 [0.058 to 0.124]
  Env-1-ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Env-1-ZM96 (Month 12) | 0.082 [0.063 to 0.119] | 0.099 [0.062 to 0.107] | 0.057 [0.042 to 0.073] | 0.09 [0.049 to 0.101]
  Env-1-ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Env-1-ZM96 (Month 12.5) | 0.127 [0.087 to 0.146] | 0.132 [0.088 to 0.144] | 0.069 [0.044 to 0.09] | 0.111 [0.088 to 0.12]
  Env-1-ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Env-1-ZM96 (Month 18) | 0.114 [0.064 to 0.127] | 0.115 [0.083 to 0.126] | 0.066 [0.039 to 0.095] | 0.085 [0.046 to 0.111]
  Env-2-ZM96 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  Env-2-ZM96 (Month 6.5) | 0.019 [0.011 to 0.05] | 0.026 [0.013 to 0.066] | 0.029 [0.014 to 0.037] | 0.023 [0.018 to 0.036]
  Env-2-ZM96 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  Env-2-ZM96 (Month 12) | 0.01 [0.001 to 0.015] | 0.026 [0.012 to 0.044] | 0.028 [0.009 to 0.042] | 0.02 [0.014 to 0.029]
  Env-2-ZM96 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  Env-2-ZM96 (Month 12.5) | 0.015 [0.006 to 0.045] | 0.039 [0.014 to 0.07] | 0.017 [0.009 to 0.034] | 0.02 [0.006 to 0.045]
  Env-2-ZM96 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  Env-2-ZM96 (Month 18) | 0.013 [0.005 to 0.019] | 0.025 [0.013 to 0.051] | 0.012 [0.008 to 0.04] | 0.022 [0.011 to 0.029]
  LAI-Gag (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  LAI-Gag (Month 6.5) | 0.051 [0.017 to 0.064] | 0.055 [0.024 to 0.072] | 0.025 [0.008 to 0.051] | 0.038 [0.031 to 0.072]
  LAI-Gag (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  LAI-Gag (Month 12) | 0.036 [0.008 to 0.055] | 0.027 [0.006 to 0.05] | 0.019 [0.007 to 0.036] | 0.027 [0.012 to 0.059]
  LAI-Gag (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  LAI-Gag (Month 12.5) | 0.031 [0.014 to 0.061] | 0.035 [0.019 to 0.058] | 0.038 [0.021 to 0.054] | 0.035 [0.009 to 0.067]
  LAI-Gag (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  LAI-Gag (Month 18) | 0.02 [0.015 to 0.039] | 0.027 [0.019 to 0.062] | 0.017 [0.006 to 0.033] | 0.035 [0.017 to 0.059]
  TV1 gp120 (Month 6.5): number analyzed (Participants) | 27 | 27 | 28 | 17
  TV1 gp120 (Month 6.5) | 0.111 [0.076 to 0.146] | 0.13 [0.095 to 0.142] | 0.108 [0.075 to 0.136] | 0.091 [0.06 to 0.122]
  TV1 gp120 (Month 12): number analyzed (Participants) | 26 | 29 | 28 | 17
  TV1 gp120 (Month 12) | 0.079 [0.056 to 0.109] | 0.111 [0.071 to 0.12] | 0.084 [0.056 to 0.115] | 0.078 [0.031 to 0.095]
  TV1 gp120 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  TV1 gp120 (Month 12.5) | 0.137 [0.094 to 0.147] | 0.146 [0.113 to 0.157] | 0.095 [0.062 to 0.129] | 0.1 [0.071 to 0.133]
  TV1 gp120 (Month 18): number analyzed (Participants) | 24 | 28 | 29 | 15
  TV1 gp120 (Month 18) | 0.109 [0.073 to 0.14] | 0.118 [0.112 to 0.135] | 0.084 [0.061 to 0.11] | 0.069 [0.035 to 0.106]

33. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C)
Description: as for outcome 1
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 29 | 32 | 16
Participants
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 30 | 28 | 31 | 16
  1086C_D7gp120.avi/293F (Month 12.5) | 30 | 27 | 31 | 16
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 29 | 29 | 30 | 16
  96ZM651.D11gp120.avi (Month 12.5) | 26 | 28 | 30 | 15
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  TV1c8_D11gp120.avi/293F (Month 12.5) | 28 | 28 | 29 | 15
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 28 | 28 | 32 | 16
  1086C_D7gp120.avi/293F (Month 18) | 27 | 27 | 32 | 16
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 27 | 29 | 31 | 15
  96ZM651.D11gp120.avi (Month 18) | 17 | 22 | 28 | 7
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  TV1c8_D11gp120.avi/293F (Month 18) | 26 | 28 | 30 | 15

34. Secondary Outcome: Level of Vaccine-induced Serum IgG Ab Binding to the 3 gp120 Env Proteins Contained in the Vaccine Regimen (ZM96, TV1.C, and 1086.C)
Description: as for outcome 22
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 28 | 32 | 16
relative fluorescence units
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 30 | 27 | 31 | 16
  1086C_D7gp120.avi/293F (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 26 | 28 | 30 | 15
  96ZM651.D11gp120.avi (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 28 | 28 | 29 | 15
  TV1c8_D11gp120.avi/293F (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 27 | 27 | 32 | 16
  1086C_D7gp120.avi/293F (Month 18) | 22000 [13447.4 to 22000] | 22000 [17031.4 to 22000] | 22000 [16465.8 to 22000] | 16187 [8260.8 to 22000]
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 17 | 22 | 28 | 7
  96ZM651.D11gp120.avi (Month 18) | 6135.8 [4058.2 to 10887] | 5439 [2617.8 to 8736.1] | 5372.6 [3140.4 to 12123.9] | 2794 [2226 to 4364.1]
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 26 | 28 | 30 | 15
  TV1c8_D11gp120.avi/293F (Month 18) | 8367.6 [2745.8 to 21097.6] | 8893.4 [3450.6 to 20507.7] | 20549 [8176.7 to 22000] | 6794.5 [2788.2 to 9961.5]

35. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG Ab Binding to V2 Env Proteins
Description: as for outcome 1
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 29 | 32 | 16
Participants
  00MSA 4076 gp140 (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  00MSA 4076 gp140 (Month 12.5) | 26 | 28 | 29 | 15
  A1.con.env03 140 CF (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  A1.con.env03 140 CF (Month 12.5) | 27 | 28 | 29 | 15
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  AE.A244 V1V2 Tags/293F (Month 12.5) | 21 | 27 | 27 | 14
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  C.1086C_V1_V2 Tags (Month 12.5) | 19 | 21 | 22 | 9
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  Con 6 gp120/B (Month 12.5) | 26 | 28 | 29 | 15
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 30 | 29 | 31 | 16
  Con S gp140 CFI (Month 12.5) | 28 | 28 | 30 | 15
  gp41 (Month 12.5): number analyzed (Participants) | 30 | 28 | 30 | 16
  gp41 (Month 12.5) | 0 | 0 | 3 | 2
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 26 | 28 | 27 | 15
  gp70-96ZM651.02 V1v2 (Month 12.5) | 10 | 18 | 18 | 7
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 16 | 25 | 24 | 9
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 28 | 28 | 28 | 16
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 12 | 22 | 23 | 8
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 27 | 28 | 28 | 16
  gp70_B.CaseA_V1_V2 (Month 12.5) | 11 | 20 | 22 | 6
  00MSA 4076 gp140 (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  00MSA 4076 gp140 (Month 18) | 11 | 12 | 18 | 4
  A1.con.env03 140 CF (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  A1.con.env03 140 CF (Month 18) | 23 | 26 | 29 | 11
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  AE.A244 V1V2 Tags/293F (Month 18) | 5 | 9 | 12 | 2
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  C.1086C_V1_V2 Tags (Month 18) | 1 | 3 | 3 | 1
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 15
  Con 6 gp120/B (Month 18) | 13 | 17 | 25 | 6
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 28 | 29 | 32 | 16
  Con S gp140 CFI (Month 18) | 25 | 28 | 31 | 15
  gp41 (Month 18): number analyzed (Participants) | 28 | 28 | 31 | 16
  gp41 (Month 18) | 0 | 1 | 3 | 1
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 25 | 28 | 28 | 14
  gp70-96ZM651.02 V1v2 (Month 18) | 1 | 3 | 4 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 26 | 28 | 29 | 15
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 4 | 10 | 11 | 1
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 27 | 28 | 29 | 15
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 1 | 3 | 7 | 1
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 26 | 28 | 29 | 15
  gp70_B.CaseA_V1_V2 (Month 18) | 1 | 2 | 6 | 1

36. Secondary Outcome: Level of Vaccine-induced Serum IgG Ab Binding to V2 Env Proteins
Description: as for outcome 22
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 30 | 28 | 32 | 16
relative fluorescence units
  00MSA 4076 gp140 (Month 12.5): number analyzed (Participants) | 26 | 28 | 29 | 15
  00MSA 4076 gp140 (Month 12.5) | 22000 [18877.6 to 22000] | 22000 [13449.4 to 22000] | 22000 [17787.8 to 22000] | 22000 [11267.2 to 22000]
  A1.con.env03 140 CF (Month 12.5): number analyzed (Participants) | 27 | 28 | 29 | 15
  A1.con.env03 140 CF (Month 12.5) | 22000 [20752 to 22000] | 22000 [17453.4 to 22000] | 22000 [22000 to 22000] | 22000 [16264.4 to 22000]
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 21 | 27 | 27 | 14
  AE.A244 V1V2 Tags/293F (Month 12.5) | 4553.5 [2286.2 to 9393.8] | 3313.8 [1245.9 to 10641.6] | 5728.8 [2011.8 to 10929.1] | 1034.2 [482.6 to 5401.9]
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 19 | 21 | 22 | 9
  C.1086C_V1_V2 Tags (Month 12.5) | 2021.2 [1142.2 to 3862.8] | 3476 [906 to 6288.5] | 3484.6 [994 to 8674.6] | 1380.2 [601 to 3883]
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 26 | 28 | 29 | 15
  Con 6 gp120/B (Month 12.5) | 22000 [22000 to 22000] | 22000 [20433.4 to 22000] | 22000 [22000 to 22000] | 22000 [15222.2 to 22000]
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 28 | 28 | 30 | 15
  Con S gp140 CFI (Month 12.5) | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  gp41 (Month 12.5): number analyzed (Participants) | 0 | 0 | 3 | 2
  gp41 (Month 12.5) |  |  | 4644.8 [3651.8 to 13322.4] | 8348.5 [5951.1 to 10745.9]
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 10 | 18 | 18 | 7
  gp70-96ZM651.02 V1v2 (Month 12.5) | 1427.2 [891.8 to 9947.6] | 3770.8 [1125 to 10077.4] | 8793.6 [1318.6 to 21615.9] | 1639.8 [1290.2 to 6055.9]
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 16 | 25 | 24 | 9
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 1407.4 [993.3 to 3027.4] | 2057.8 [714.5 to 6260.2] | 12436.5 [1806.4 to 22000] | 2031.8 [1158.8 to 4055.5]
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 12 | 22 | 23 | 8
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 1213.2 [734.6 to 3588.6] | 2332.9 [732.9 to 5249.1] | 8987.2 [2613.6 to 22000] | 1324.4 [941.3 to 3481.6]
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 11 | 20 | 22 | 6
  gp70_B.CaseA_V1_V2 (Month 12.5) | 763.5 [670.1 to 3615.2] | 2246.5 [999.1 to 5417.9] | 8372.5 [1587.8 to 21441.9] | 2869.5 [1171.8 to 4368.3]
  00MSA 4076 gp140 (Month 18): number analyzed (Participants) | 11 | 12 | 18 | 4
  00MSA 4076 gp140 (Month 18) | 1954 [1242.2 to 3022] | 2546.9 [1072.2 to 7260.1] | 1571 [1131.2 to 3575.8] | 1351.9 [1189.6 to 1367.8]
  A1.con.env03 140 CF (Month 18): number analyzed (Participants) | 23 | 26 | 29 | 11
  A1.con.env03 140 CF (Month 18) | 1106 [444.2 to 2628] | 1552.5 [607 to 3231.8] | 1853.2 [929.5 to 4194.5] | 961.5 [695.8 to 1429.6]
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 5 | 9 | 12 | 2
  AE.A244 V1V2 Tags/293F (Month 18) | 137 [110.2 to 484] | 462 [371.2 to 512.5] | 362.2 [194.8 to 1003.6] | 445.9 [429.3 to 462.4]
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 1 | 3 | 3 | 1
  C.1086C_V1_V2 Tags (Month 18) | 1204.5 [1204.5 to 1204.5] | 1523.2 [1067.4 to 5288.9] | 821.8 [714.1 to 2419.4] | 909 [909 to 909]
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 13 | 17 | 25 | 6
  Con 6 gp120/B (Month 18) | 2373.2 [1574 to 4438.2] | 2805 [1459.5 to 4348.8] | 2405.5 [1517.5 to 4459.5] | 1185.2 [993.6 to 1463.2]
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 25 | 28 | 31 | 15
  Con S gp140 CFI (Month 18) | 8793.8 [3178.8 to 16947.8] | 9031.1 [3772.2 to 22000] | 13261.8 [7458.2 to 22000] | 5032.5 [3082 to 9318.4]
  gp41 (Month 18): number analyzed (Participants) | 0 | 1 | 3 | 1
  gp41 (Month 18) |  | 2549.2 [2549.2 to 2549.2] | 7284.8 [5785.5 to 14642.4] | 19096.5 [19096.5 to 19096.5]
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 1 | 3 | 4 | 1
  gp70-96ZM651.02 V1v2 (Month 18) | 370.8 [370.8 to 370.8] | 584 [541.4 to 872.1] | 987.8 [590.4 to 1672.9] | 2221.8 [2221.8 to 2221.8]
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 4 | 10 | 11 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 163.1 [125.2 to 272.5] | 180.2 [130.4 to 208.4] | 1319.2 [605.5 to 1729.8] | 1114.2 [1114.2 to 1114.2]
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 1 | 3 | 7 | 1
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 244.5 [244.5 to 244.5] | 1593.8 [914.8 to 1638.4] | 1332 [425 to 1556] | 1227.5 [1227.5 to 1227.5]
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 1 | 2 | 6 | 1
  gp70_B.CaseA_V1_V2 (Month 18) | 314.2 [314.2 to 314.2] | 1717.6 [1210.9 to 2224.3] | 623.8 [383.3 to 886.9] | 593.2 [593.2 to 593.2]

37. Secondary Outcome: Occurrence of Vaccine-induced Serum IgG3 Ab Binding to Env Proteins
Description: as for outcome 27
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 31 | 29 | 32 | 17
Participants
  1086C_D7gp120.avi/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  1086C_D7gp120.avi/293F (Month 12.5) | 28 | 28 | 29 | 15
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  96ZM651.D11gp120.avi (Month 12.5) | 14 | 17 | 14 | 8
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 16
  AE.A244 V1V2 Tags/293F (Month 12.5) | 6 | 9 | 13 | 4
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 16
  C.1086C_V1_V2 Tags (Month 12.5) | 4 | 7 | 10 | 1
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  Con 6 gp120/B (Month 12.5) | 6 | 10 | 5 | 4
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  Con S gp140 CFI (Month 12.5) | 18 | 21 | 19 | 10
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 31 | 17
  TV1c8_D11gp120.avi/293F (Month 12.5) | 25 | 25 | 28 | 13
  gp41 (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 16
  gp41 (Month 12.5) | 0 | 0 | 0 | 1
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 30 | 29 | 29 | 15
  gp70-96ZM651.02 V1v2 (Month 12.5) | 3 | 3 | 5 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 2 | 2 | 8 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 1 | 2 | 7 | 0
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 31 | 29 | 30 | 15
  gp70_B.CaseA_V1_V2 (Month 12.5) | 1 | 2 | 4 | 0
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  1086C_D7gp120.avi/293F (Month 18) | 11 | 16 | 15 | 4
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  96ZM651.D11gp120.avi (Month 18) | 0 | 0 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 15
  AE.A244 V1V2 Tags/293F (Month 18) | 1 | 0 | 5 | 0
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 15
  C.1086C_V1_V2 Tags (Month 18) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  Con 6 gp120/B (Month 18) | 0 | 0 | 1 | 0
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  Con S gp140 CFI (Month 18) | 4 | 4 | 0 | 0
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 29 | 29 | 32 | 16
  TV1c8_D11gp120.avi/293F (Month 18) | 6 | 6 | 4 | 2
  gp41 (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 15
  gp41 (Month 18) | 0 | 0 | 0 | 2
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 28 | 29 | 30 | 14
  gp70-96ZM651.02 V1v2 (Month 18) | 1 | 0 | 2 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 1 | 0 | 1 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 1 | 0 | 1 | 0
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 29 | 29 | 31 | 14
  gp70_B.CaseA_V1_V2 (Month 18) | 1 | 0 | 0 | 0

38. Secondary Outcome: Level of Vaccine-induced Serum IgG3 Ab Binding to Env Proteins
Description: as for outcome 28
Time Frame: Measured at Months 12.5 and 18.
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
Number analyzed (Participants) | 28 | 28 | 29 | 15
relative fluorescence units
  1086C_D7gp120.avi/293F (Month 12.5) | 1049.2 [390 to 2565.1] | 1184.2 [711.1 to 3716.6] | 1086.2 [606.8 to 2699.8] | 1739 [593.4 to 5582.2]
  96ZM651.D11gp120.avi (Month 12.5): number analyzed (Participants) | 14 | 17 | 14 | 8
  96ZM651.D11gp120.avi (Month 12.5) | 300.9 [161.9 to 838.8] | 314.5 [149 to 681.5] | 314.9 [189.6 to 439.3] | 264.5 [203.9 to 391]
  AE.A244 V1V2 Tags/293F (Month 12.5): number analyzed (Participants) | 6 | 9 | 13 | 4
  AE.A244 V1V2 Tags/293F (Month 12.5) | 283.9 [178.3 to 762] | 271 [193.5 to 666.2] | 480 [289.2 to 697] | 479.1 [308.5 to 5950.9]
  C.1086C_V1_V2 Tags (Month 12.5): number analyzed (Participants) | 4 | 7 | 10 | 1
  C.1086C_V1_V2 Tags (Month 12.5) | 470 [320.7 to 1060.8] | 197.8 [152.6 to 332.5] | 379.2 [218.2 to 473] | 22000 [22000 to 22000]
  Con 6 gp120/B (Month 12.5): number analyzed (Participants) | 6 | 10 | 5 | 4
  Con 6 gp120/B (Month 12.5) | 284 [197.3 to 345.2] | 329.5 [174.1 to 376] | 540 [278.5 to 672.5] | 203 [131 to 510.4]
  Con S gp140 CFI (Month 12.5): number analyzed (Participants) | 18 | 21 | 19 | 10
  Con S gp140 CFI (Month 12.5) | 264.1 [179 to 623.1] | 322.8 [202.2 to 1225.2] | 208.2 [160.5 to 382.6] | 476.8 [118.7 to 581.4]
  TV1c8_D11gp120.avi/293F (Month 12.5): number analyzed (Participants) | 25 | 25 | 28 | 13
  TV1c8_D11gp120.avi/293F (Month 12.5) | 586.8 [385.5 to 2959.5] | 673.8 [415 to 2072.2] | 439.4 [199.9 to 1111.1] | 1017.2 [708 to 3056.2]
  gp41 (Month 12.5): number analyzed (Participants) | 0 | 0 | 0 | 1
  gp41 (Month 12.5) |  |  |  | 3020.8 [3020.8 to 3020.8]
  gp70-96ZM651.02 V1v2 (Month 12.5): number analyzed (Participants) | 3 | 3 | 5 | 1
  gp70-96ZM651.02 V1v2 (Month 12.5) | 157.8 [130.9 to 992.2] | 354 [287.8 to 431.9] | 2402.8 [1323.5 to 3308.5] | 4707.5 [4707.5 to 4707.5]
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 2 | 2 | 8 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 853.5 [564.1 to 1142.9] | 231.6 [181.9 to 281.3] | 487.8 [167.2 to 1114.6] |
  gp70_B.CaseA2 V1/V2/169K (Month 12.5): number analyzed (Participants) | 1 | 2 | 7 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 12.5) | 2010.8 [2010.8 to 2010.8] | 255.4 [191.4 to 319.3] | 551 [175 to 850.4] |
  gp70_B.CaseA_V1_V2 (Month 12.5): number analyzed (Participants) | 1 | 2 | 4 | 0
  gp70_B.CaseA_V1_V2 (Month 12.5) | 1262.5 [1262.5 to 1262.5] | 233.5 [205.1 to 261.9] | 1457.8 [642 to 2307.9] |
  1086C_D7gp120.avi/293F (Month 18): number analyzed (Participants) | 11 | 16 | 15 | 4
  1086C_D7gp120.avi/293F (Month 18) | 204 [146.2 to 522.4] | 266.4 [172.9 to 555.9] | 167.5 [158.5 to 217.5] | 133 [109.4 to 236.1]
  96ZM651.D11gp120.avi (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 0
  AE.A244 V1V2 Tags/293F (Month 18): number analyzed (Participants) | 1 | 0 | 5 | 0
  AE.A244 V1V2 Tags/293F (Month 18) | 187.8 [187.8 to 187.8] |  | 245.2 [197.2 to 479.5] |
  C.1086C_V1_V2 Tags (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 0
  Con 6 gp120/B (Month 18): number analyzed (Participants) | 0 | 0 | 1 | 0
  Con 6 gp120/B (Month 18) |  |  | 368.8 [368.8 to 368.8] |
  Con S gp140 CFI (Month 18): number analyzed (Participants) | 4 | 4 | 0 | 0
  Con S gp140 CFI (Month 18) | 126.6 [100 to 155.2] | 136.6 [126.4 to 156.8] |  |
  TV1c8_D11gp120.avi/293F (Month 18): number analyzed (Participants) | 6 | 6 | 4 | 2
  TV1c8_D11gp120.avi/293F (Month 18) | 451.2 [202.6 to 915.9] | 198.9 [125.4 to 362] | 725.9 [239.6 to 1298.6] | 6535.8 [3329.8 to 9741.8]
  gp41 (Month 18): number analyzed (Participants) | 0 | 0 | 0 | 2
  gp41 (Month 18) |  |  |  | 9170.6 [6114.3 to 12226.9]
  gp70-96ZM651.02 V1v2 (Month 18): number analyzed (Participants) | 1 | 0 | 2 | 0
  gp70-96ZM651.02 V1v2 (Month 18) | 434.8 [434.8 to 434.8] |  | 196.6 [151.1 to 242.2] |
  gp70-TV1.GSKvacV1V2/293F (Month 18): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 18) | 534.8 [534.8 to 534.8] |  | 170.5 [170.5 to 170.5] |
  gp70_B.CaseA2 V1/V2/169K (Month 18): number analyzed (Participants) | 1 | 0 | 1 | 0
  gp70_B.CaseA2 V1/V2/169K (Month 18) | 887.5 [887.5 to 887.5] |  | 177.5 [177.5 to 177.5] |
  gp70_B.CaseA_V1_V2 (Month 18): number analyzed (Participants) | 1 | 0 | 0 | 0
  gp70_B.CaseA_V1_V2 (Month 18) | 474 [474 to 474] |  |  |

ADVERSE EVENTS:
Time Frame: Serious adverse events, adverse events of special interest, and new chronic conditions requiring medical intervention of more than 30 days were collected through month 18. All other AEs were collected through 30 days after each vaccination (vaccinations were given at months 0, 1, 3, and 6 for Groups 1, 2, and 4 and at months 0, 1, and 6 for Group 3).
Description: Adverse events of special interest were described in Appendix N of the protocol. AESI for this protocol include but are not limited to potential immune-mediated diseases.
Arm/Group | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/36 | 0/36 | 1/24
Other Adverse Events (participants affected / at risk) | 28/36 | 28/36 | 26/36 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) (N=36) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) (N=36) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) (N=36) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12) (N=24)
Any Event in SOC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120/MF59 mo(3,6,12) (N=36) | Group 2: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120+Alum mo(3,6,12) (N=36) | Group 3: ALVAC mo(0,1,6,12) + Bivalent Subtype C gp120/MF59 mo(0,1,6,12) (N=36) | Group 4: ALVAC mo(0,1,3,6,12) + Bivalent Subtype C gp120 mo(3,6,12) (N=24)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 4 (4) | 4 (6) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 15 (29) | 14 (26) | 10 (16) | 11 (16)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (4)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 4 (5) | 5 (8) | 2 (4) | 0 (0)
Genitourinary tract gonococcal infection (Infections and infestations) | 2 (3) | 1 (2) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (6) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 4 (4) | 3 (5)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 20 (35) | 14 (26) | 10 (17) | 6 (10)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (4) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 4 (5) | 2 (4)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 10 (17) | 6 (8) | 4 (5) | 2 (2)
Blood pressure increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 5 (6) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (5) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 2 (2) | 6 (7) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 2 (3) | 2 (3) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Any Event in SOC (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5) | 4 (4) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03284710/Prot_SAP_000.pdf